CLINICAL TRIAL: NCT03287245
Title: A Phase II, Single-Arm, Open-Label Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Idasanutlin Monotherapy in Patients With Hydroxyurea-Resistant/Intolerant Polycythemia Vera
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Idasanutlin Monotherapy in Participants With Hydroxyurea-Resistant/Intolerant Polycythemia Vera
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue the development of idasanutlin in the polycythemia vera indication.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP39761; 2017-000861-58 (EudraCT Number)
Record Dates: First submitted 2017-09-08; First posted 2017-09-19 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Polycythemia Vera
Keywords: polycythemia vera; PV; P vera; myeloproliferative diseases; hematologic diseases; myeloproliferative neoplasm; MPN
MeSH Terms: conditions — Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders | interventions — RG7388

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idasanutlin (Experimental): Two cohorts of ruxolitinib-naïve and ruxolitinib-resitant or intolerant participants will be enrolled to receive idasanutlin once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
  Interventions: Drug: Idasanutlin

INTERVENTIONS:
Drug: Idasanutlin — All participants will receive 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years). Intra-participant dose-escalation to 200 mg daily for 5 days may be permitted after Cycle 3 for those who demonstrate no hematocrit (Hct) control and/or for those with inadequately controlled leukocytosis and/or thrombocytosis in which the investigator judges that better control is important.
  Other Names: RO5503781; RG7388

SUMMARY:
This is an open-label, single-arm study of idasanutlin monotherapy in participants with hydroxyurea (HU)-resistant/intolerant Polycythemia vera (PV). The study will include two phases: initial phase and expansion phase. The initial phase will assess the safety and efficacy of idasanutlin monotherapy in ruxolitinib naïve and ruxolitinib-resistant or intolerant patients, respectively. If the initial phase shows promising results for ruxolitinib-resistant or intolerant patients, an expansion phase will be opened to further characterize the efficacy of idasanutlin.

ELIGIBILITY:
Inclusion Criteria:

* Documentation that the participant has met the revised 2016 World Health Organization (WHO) criteria for the diagnosis of polycythemia vera (PV)
* Hematocrit at screening and at initiation of idasanutlin greater than (>)40%
* Phlebotomy-dependent participants with splenomegaly by magnetic resonance imaging (MRI) or computerized tomography (CT) imaging (greater than or equal to [≥]450 cubic centimeters [cm^3]) or without splenomegaly (less than [<]450 cm^3 or prior splenectomy)
* Resistance to/intolerance to hydroxyurea according to modified European Leukemia Net (ELN) criteria
* For participants in the ruxolitinib intolerant or resistant group, in addition to previous hydroxyurea intolerance/resistance: Therapy-resistant PV after at least 6 months of treatment with ruxolitinib, as defined in the protocol; Ruxolitinib intolerance, as defined in the protocol; and Documentation of adverse events likely caused by ruxolitinib (assessment of attending physician) and that are of a severity that preclude further treatment with ruxolitinib (as per judgment of the attending physician and the patient)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participants must be willing to submit the blood sampling and bone marrow sampling for the pharmacokinetic (PK) and pharmacodynamic analyses and exploratory biomarkers
* Adequate hepatic and renal function
* Ability and willingness to comply with the study protocol procedures, including clinical outcome assessment measures
* For women of childbearing potential: agreement to use contraceptive methods that result in a failure rate of less than (<)1% per year during the treatment period and for at least 6 weeks after the last dose of idasanutlin
* For men: Agreement to use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for at least 90 days after the last dose of idasanutlin

Exclusion Criteria:

* Meets the criteria for post-PV myelofibrosis as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT)
* Blast phase disease (>20% blasts in the marrow or peripheral blood)
* Clinically-significant thrombosis within 3 months of screening
* Participants who must receive CYP2C8 inhibitors, substrates and inducers, strong CYP3A4 inducers, or OATP1B1/3 substrates while on study. These must be discontinued 7 days (inhibitors and substrates) or 14 days (inducers) prior to start of study medication
* Previously treated with murine double minute 2 (MDM2) antagonist therapies or receiving interferon-alpha, anagrelide, or ruxolitinib within 28 days or 5 half-lives (whichever is shorter), or hydroxyurea within 1 day, or receiving any other cytoreductive or investigational agents within 28 days or 5 half-lives (whichever is shorter) of initial dose. Aspirin is permitted per treatment guidelines for PV unless medically contraindicated
* Patients with evidence of electrolyte imbalance such as hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypomagnesemia, and hypermagnesemia of Grade >1 intensity, as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0, prior to dosing on Cycle 1 Day 1. Treatment for correction of electrolyte imbalances is permitted to meet eligibility
* Neutrophil count <1.5 × 10^9/Liter (L) prior to dosing on Cycle 1 Day 1
* Platelet count less than or equal to (≤)150 × 10^9/L prior to dosing on Cycle 1 Day 1
* Women who are pregnant or breastfeeding
* Ongoing serious non-healing wound, ulcer, or bone fracture
* History of major organ transplant
* Uncontrolled intercurrent illness including, but not limited to hepatitis, concurrent malignancy that could affect compliance with the protocol or interpretation of results, hepatitis A, B, and C, human immunodeficiency virus (HIV)-positive, ongoing or active infection, clinically significant cardiac disease (New York Heart Association Class III or IV), symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Concurrent malignancy exceptions include: Curatively treated carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal- or squamous-cell skin cancer, Stage I melanoma, or low-grade, early-stage localized prostate cancer. Any previously treated early-stage non-hematological malignancy that has been in remission for at least 2 years is also permitted.
* Patients with active gastrointestinal conditions (Crohn's disease, ulcerative colitis, diverticulosis associated colitis, and Behçet's disease)
* Clinically significant toxicity (other than alopecia) from prior therapy that has not resolved to Grade ≤1 (according to the NCI CTCAE, v4.0) prior to Cycle 1 Day 1
* Cardiovascular disease, such as: uncontrolled arterial hypertension; symptomatic congestive heart failure or ejection fraction below 55% at screening, or left ventricular hypertrophy; any significant structural abnormality of the heart at screening echocardiogram; unstable angina pectoris; presence or history of any type of supraventricular and ventricular arrhythmias, including lone atrial fibrillation or flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (5):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of Kansas Cancer Center; Westwood Cancer Center/BMT Output Clinic, Kansas City, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - University of Texas Health Sciences Center in San Antonio, San Antonio, Texas
- Australia (2):
  - Royal Adelaide Hospital; Haematology Clinical Trials, Adelaide, South Australia
  - Peter MacCallum Cancer Centre; Department of Haematology, Melbourne, Victoria
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Italy (3):
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi; Ematologia, Varese, Lombardy
  - Az. Ospedaliero-Universitaria Careggi; CRIMM, Florence, Tuscany

REFERENCES:
- [Derived] Mascarenhas J, Passamonti F, Burbury K, El-Galaly TC, Gerds A, Gupta V, Higgins B, Wonde K, Jamois C, Kovic B, Huw LY, Katakam S, Maffioli M, Mesa R, Palmer J, Bellini M, Ross DM, Vannucchi AM, Yacoub A. The MDM2 antagonist idasanutlin in patients with polycythemia vera: results from a single-arm phase 2 study. Blood Adv. 2022 Feb 22;6(4):1162-1174. doi: 10.1182/bloodadvances.2021006043. PMID 34933330
- See also: Pioneeringhealthcare.com supports an online community of people impacted by Polycythemia Vera (PV, or P Vera), and provides explanations of medical terms and insights about the purpose of Roche's new clinical trial (NP39761) for patients with P Vera. — https://www.pioneeringhealthcare.com/p-vera

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants were screened for enrollment; 21 were failed screening. 27 were enrolled and received study treatment. All 27 patients were discontinued from study before the planned date of follow-up.
Groups:
- Ruxolitinib-naïve Participants With Splenomegaly; Ruxolitinib-naïve Participants Without Splenomegaly; Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly; Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Period: Overall Study
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Started | 15 | 5 | 6 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 5 | 6 | 1
Not completed — Study terminated by sponsor | 3 | 0 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 3 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly | Total
Number analyzed (Participants) | 15 | 5 | 6 | 1 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (10.7) | 56.8 (8.8) | 60.3 (8.4) | 55 (0) | 56.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 0 | 11
  Male | 13 | 0 | 2 | 1 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 5 | 6 | 1 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 1
  White | 14 | 5 | 6 | 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ruxolitinib-Naïve Participants With Splenomegaly at Baseline Who Achieved Composite Response at Week 32
Description: Composite response is defined as hematocrit (Hct) control without phlebotomy and ≥35% decrease in spleen size by imaging at Week 32. Hct control is defined as protocol-specified ineligibility for phlebotomy between Weeks 8 to 32 and ≤1 instance of phlebotomy eligibility between first dose and Week 8. Eligibility for phlebotomy is defined as a Hct of ≥45% that was ≥3% higher than baseline level or a Hct of >48%. One Cycle is 28 Days.
Time Frame: Week 32
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly
Number analyzed (Participants) | 9
Percentage of Participants | 44.4

2. Primary Outcome: Percentage of Ruxolitinib-Naïve Participants Without Splenomegaly at Baseline Who Achieved Hematocrit (Hct) Control Without Phlebotomy at Week 32
Description: Hct control is defined as protocol-specified ineligibility for phlebotomy between Weeks 8 to 32 and ≤1 instance of phlebotomy eligibility between first dose and Week 8. Eligibility for phlebotomy is defined as a Hct level ≥45% that was ≥3% higher than baseline level or a Hct level of >48%.
Time Frame: Week 32
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants Without Splenomegaly
Number analyzed (Participants) | 2
Percentage of Participants | 100

3. Primary Outcome: Percentage of All Ruxolitinib-Naïve Participants (Irrespective of Spleen Size) Who Achieved Hct Control Without Phlebotomy at Week 32
Description: as for outcome 2
Time Frame: Week 32
Population: ITT population
Measure: Number; unit: Percentage of Participants
Groups:
- Total Ruxolitinib-Naïve Participants: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Naïve Participants Without Splenomegaly | Total Ruxolitinib-Naïve Participants
Number analyzed (Participants) | 9 | 2 | 11
Percentage of Participants | 44.4 | 100 | 54.5

4. Primary Outcome: Percentage of All Ruxolitinib-Resistant or Intolerant Participants Who Achieved Hct Control Without Phlebotomy at Week 32
Description: as for outcome 2
Time Frame: From Baseline to Week 32 (Cycle 8 Day 28)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Groups:
- Total Ruxolitinib-Resistant or Intolerant Participants: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years)
Arm/Group | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly | Total Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 4 | 1 | 5
Percentage of Participants | 75.0 | 0 | 60

5. Secondary Outcome: Percentage of All Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants Who Achieved Complete Hematologic Response at Week 32
Description: Complete hematologic response requires all of the following: Hct control without phlebotomy; White blood cell (WBC) count ≤10 × 10^9/Liter (L) at Week 32; and Platelet count ≤400 × 10^9/L at Week 32. Hct control is defined as protocol-specified ineligibility for phlebotomy between Weeks 8 to 32 and ≤1 instance of phlebotomy eligibility between first dose and Week 8. Eligibility for phlebotomy is defined as a Hct level ≥45% that was ≥3% higher than baseline level or a Hct level of >48%.
Time Frame: Week 32 (Cycle 8 Day 28)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 9 | 2 | 4 | 1
Percentage of Participants | 33.3 | 100 | 75.0 | 0

6. Secondary Outcome: Percentage of All Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants Who Achieved Complete Hematologic Remission at Cycle 11 Day 28
Description: Complete hematologic remission requires all of the following: Hct control without phlebotomy between Weeks 32 and Cycle 11 Day 28; WBC count ≤10 × 10^9/L at Cycle 11 Day 28; and Platelet count ≤400 × 10^9/L at Week 32. Hct control is defined as protocol-specified ineligibility for phlebotomy. Eligibility for phlebotomy is defined as a Hct level ≥45% that was ≥3% higher than baseline level or a Hct level of >48%.
Time Frame: Cycle 11 Day 28
Population: ITT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 5 | 1 | 1 | 1
Percentage of Participants | 40 | 100 | 0 | 0

7. Secondary Outcome: Duration of Complete Hematologic Remission, With a Durable Responder Defined as a Participant in Remission at Week 32 and Cycle 11 Day 28
Description: Complete hematologic remission requires all of the following: Hct control without phlebotomy between Week 32 (Cycle 8 Day 28) and Cycle 11 Day 28; WBC count ≤10 × 10^9/L at Cycle 11 Day 28; and Platelet count ≤400 × 10^9/L at Week 32. Hct control is defined as protocol-specified ineligibility for phlebotomy. Eligibility for phlebotomy is defined as a Hct level ≥45% that was ≥3% higher than baseline level or a Hct level of >48%
Time Frame: Week 32 (Cycle 8 Day 28), Cycle 11 Day 28
Population: ITT population. The "number of participants analyzed" is the number of patients (total n) per arm. "The number analyzed" was the number of patients evaluable at that specific timepoint. Not all participants of each arm were evaluable at each time point.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Participants
  Cycle 11, Day 28: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 11, Day 28 | 2 | 1 | 0 | 0
  Week 32: number analyzed (Participants) | 9 | 2 | 4 | 1
  Week 32 | 3 | 2 | 3 | 0

8. Secondary Outcome: Percentage of Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly at Baseline by Response Per Modified European Leukemia Net (ELN) Criteria
Description: Complete response (CR) includes all of the following: Hct <45% without phlebotomy; Platelet count ≤400 × 10^9/L; WBC count ≤10 × 10^9/L; Normal spleen size on imaging; and No disease-related symptoms. Partial response (PR): in participants who do not fulfill the criteria for CR: Hct <45% without phlebotomy or response in 3 or more of the other criteria. No response (NR): any response that does not satisfy partial response. Progressive disease (PD): increased bone marrow fibrosis from baseline, and/or transformation to myelofibrosis (MF), myelodysplastic syndrome (MDS) or acute leukemia.
  All responders of each category grouped per timepoint include all categories mentioned above. There were no PD responses at any timepoint.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the end of study.
Time Frame: Baseline, Day 28 of Cycles 3, 5, 8, 11, 12, 14, 17, 20 and Final visit (28 days after post-last dose)
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly
Number analyzed (Participants) | 15 | 6
Percentage of Participants
  Baseline Complete Response | 0 | 0
  Baseline Partial Response | 0 | 0
  Baseline Progressive Disease | 0 | 0
  Baseline No Response | 0 | 0
  Cycle 3, Day 28 Complete Response | 0 | 33.3
  Cycle 3, Day 28 Partial Response | 73.3 | 50.0
  Cycle 3, Day 28 Progressive Disease | 0 | 0
  Cycle 3, Day 28 No Response | 26.7 | 16.7
  Cycle 5, Day 28 Complete Response: number analyzed (Participants) | 13 | 5
  Cycle 5, Day 28 Complete Response | 0 | 0
  Cycle 5, Day 28 Partial Response: number analyzed (Participants) | 13 | 5
  Cycle 5, Day 28 Partial Response | 76.9 | 80.0
  Cycle 5, Day 28 Progressive Disease: number analyzed (Participants) | 13 | 5
  Cycle 5, Day 28 Progressive Disease | 0 | 0
  Cycle 5, Day 28 No Response: number analyzed (Participants) | 13 | 5
  Cycle 5, Day 28 No Response | 23.1 | 20.0
  Cycle 8, Day 28 (Week 32) Complete Response: number analyzed (Participants) | 9 | 4
  Cycle 8, Day 28 (Week 32) Complete Response | 0 | 25.0
  Cycle 8, Day 28 (Week 32) Partial Response: number analyzed (Participants) | 9 | 4
  Cycle 8, Day 28 (Week 32) Partial Response | 66.7 | 50.0
  Cycle 8, Day 28 (Week 32) Progressive Disease: number analyzed (Participants) | 9 | 4
  Cycle 8, Day 28 (Week 32) Progressive Disease | 0 | 0
  Cycle 8, Day 28 (Week 32) No Response: number analyzed (Participants) | 9 | 4
  Cycle 8, Day 28 (Week 32) No Response | 33.3 | 25.0
  Cycle 11, Day 28 Complete Response: number analyzed (Participants) | 5 | 1
  Cycle 11, Day 28 Complete Response | 0 | 0
  Cycle 11, Day 28 Partial Response: number analyzed (Participants) | 5 | 1
  Cycle 11, Day 28 Partial Response | 80.0 | 100.0
  Cycle 11, Day 28 Progressive Disease: number analyzed (Participants) | 5 | 1
  Cycle 11, Day 28 Progressive Disease | 0 | 0
  Cycle 11, Day 28 No Response: number analyzed (Participants) | 5 | 1
  Cycle 11, Day 28 No Response | 20.0 | 0
  Cycle 12, Day 28 Complete Response: number analyzed (Participants) | 0 | 1
  Cycle 12, Day 28 Complete Response |  | 0
  Cycle 12, Day 28 Partial Response: number analyzed (Participants) | 0 | 1
  Cycle 12, Day 28 Partial Response |  | 0
  Cycle 12, Day 28 Progressive Disease: number analyzed (Participants) | 0 | 1
  Cycle 12, Day 28 Progressive Disease |  | 0
  Cycle 12, Day 28 No Response: number analyzed (Participants) | 0 | 1
  Cycle 12, Day 28 No Response |  | 0
  Cycle 14, Day 28 Complete Response: number analyzed (Participants) | 5 | 1
  Cycle 14, Day 28 Complete Response | 0 | 0
  Cycle 14, Day 28 Partial Response: number analyzed (Participants) | 5 | 1
  Cycle 14, Day 28 Partial Response | 80 | 100
  Cycle 14, Day 28 Progressive Disease: number analyzed (Participants) | 5 | 1
  Cycle 14, Day 28 Progressive Disease | 0 | 0
  Cycle 14, Day 28 No Response: number analyzed (Participants) | 5 | 1
  Cycle 14, Day 28 No Response | 20 | 0
  Cycle 17, Day 28 Complete Response: number analyzed (Participants) | 3 | 1
  Cycle 17, Day 28 Complete Response | 0 | 0
  Cycle 17, Day 28 Partial Response: number analyzed (Participants) | 3 | 1
  Cycle 17, Day 28 Partial Response | 33.3 | 0
  Cycle 17, Day 28 Progressive Disease: number analyzed (Participants) | 3 | 1
  Cycle 17, Day 28 Progressive Disease | 0 | 0
  Cycle 17, Day 28 No Response: number analyzed (Participants) | 3 | 1
  Cycle 17, Day 28 No Response | 66.7 | 100
  Cycle 20, Day 28 Complete Response: number analyzed (Participants) | 1 | 0
  Cycle 20, Day 28 Complete Response | 0 |
  Cycle 20, Day 28 Partial Response: number analyzed (Participants) | 1 | 0
  Cycle 20, Day 28 Partial Response | 100 |
  Cycle 20, Day 28 Progressive Disease: number analyzed (Participants) | 1 | 0
  Cycle 20, Day 28 Progressive Disease | 0 |
  Cycle 20, Day 28 No Response: number analyzed (Participants) | 1 | 0
  Cycle 20, Day 28 No Response | 0 |
  Final Visit (28 Days post-last dose) Complete Response: number analyzed (Participants) | 10 | 3
  Final Visit (28 Days post-last dose) Complete Response | 0 | 0
  Final Visit (28 Days post-last dose) Partial Response: number analyzed (Participants) | 10 | 3
  Final Visit (28 Days post-last dose) Partial Response | 20.0 | 33.3
  Final Visit (28 Days post-last dose) Progressive Disease: number analyzed (Participants) | 10 | 3
  Final Visit (28 Days post-last dose) Progressive Disease | 0 | 0
  Final Visit (28 Days post-last dose) No Response: number analyzed (Participants) | 10 | 3
  Final Visit (28 Days post-last dose) No Response | 80 | 66.7

9. Secondary Outcome: Percentage of Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly at Baseline by Response Per Modified ELN Criteria
Description: as for outcome 8
Time Frame: Baseline, Day 28 of Cycles 3, 5, 8, 11, 12, 14, 17, 20 and Final visit (28 days after post-last dose)
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 5 | 1
Percentage of Participants
  Baseline Complete Response | 0 | 0
  Baseline Partial Response | 0 | 0
  Baseline Progressive Disease | 0 | 0
  Baseline No Response | 0 | 0
  Cycle 3, Day 28 Complete Response: number analyzed (Participants) | 4 | 1
  Cycle 3, Day 28 Complete Response | 50 | 0
  Cycle 3, Day 28 Partial Response: number analyzed (Participants) | 4 | 1
  Cycle 3, Day 28 Partial Response | 50 | 0
  Cycle 3, Day 28 Progressive Disease: number analyzed (Participants) | 4 | 1
  Cycle 3, Day 28 Progressive Disease | 0 | 0
  Cycle 3, Day 28 No Response: number analyzed (Participants) | 4 | 1
  Cycle 3, Day 28 No Response | 0 | 100
  Cycle 5 Day 28 Complete Response: number analyzed (Participants) | 3 | 1
  Cycle 5 Day 28 Complete Response | 66.7 | 0
  Cycle 5 Day 28 Partial Response: number analyzed (Participants) | 3 | 1
  Cycle 5 Day 28 Partial Response | 33.3 | 0
  Cycle 5 Day 28 Progressive Disease: number analyzed (Participants) | 3 | 1
  Cycle 5 Day 28 Progressive Disease | 0 | 0
  Cycle 5 Day 28 No Response: number analyzed (Participants) | 3 | 1
  Cycle 5 Day 28 No Response | 0 | 100
  Cycle 8, Day 28 (Week 32) Complete Response: number analyzed (Participants) | 2 | 1
  Cycle 8, Day 28 (Week 32) Complete Response | 100 | 0
  Cycle 8, Day 28 (Week 32) Partial Response: number analyzed (Participants) | 2 | 1
  Cycle 8, Day 28 (Week 32) Partial Response | 0 | 0
  Cycle 8, Day 28 (Week 32) Progressive Disease: number analyzed (Participants) | 2 | 1
  Cycle 8, Day 28 (Week 32) Progressive Disease | 0 | 0
  Cycle 8, Day 28 (Week 32) No Response: number analyzed (Participants) | 2 | 1
  Cycle 8, Day 28 (Week 32) No Response | 0 | 100
  Cycle 11, day 28 Complete Response: number analyzed (Participants) | 1 | 1
  Cycle 11, day 28 Complete Response | 100 | 0
  Cycle 11, day 28 Partial Response: number analyzed (Participants) | 1 | 1
  Cycle 11, day 28 Partial Response | 0 | 0
  Cycle 11, day 28 Progressive Disease: number analyzed (Participants) | 1 | 1
  Cycle 11, day 28 Progressive Disease | 0 | 0
  Cycle 11, day 28 No Response: number analyzed (Participants) | 1 | 1
  Cycle 11, day 28 No Response | 0 | 100
  Cycle 12, Day 28 Complete Response: number analyzed (Participants) | 0 | 0
  Cycle 12, Day 28 Partial Response: number analyzed (Participants) | 0 | 0
  Cycle 12, Day 28 Progressive Disease: number analyzed (Participants) | 0 | 0
  Cycle 12, Day 28 No Response: number analyzed (Participants) | 0 | 0
  Cycle 14, Day 28 Complete Response: number analyzed (Participants) | 1 | 1
  Cycle 14, Day 28 Complete Response | 100 | 0
  Cycle 14, Day 28 Partial Response: number analyzed (Participants) | 1 | 1
  Cycle 14, Day 28 Partial Response | 0 | 0
  Cycle 14, Day 28 Progressive Disease: number analyzed (Participants) | 1 | 1
  Cycle 14, Day 28 Progressive Disease | 0 | 0
  Cycle 14, Day 28 No Response: number analyzed (Participants) | 1 | 1
  Cycle 14, Day 28 No Response | 0 | 100
  Cycle 17, Day 28 Complete Response: number analyzed (Participants) | 1 | 1
  Cycle 17, Day 28 Complete Response | 100 | 0
  Cycle 17, Day 28 Partial Response: number analyzed (Participants) | 1 | 1
  Cycle 17, Day 28 Partial Response | 0 | 0
  Cycle 17, Day 28 Progressive Disease: number analyzed (Participants) | 1 | 1
  Cycle 17, Day 28 Progressive Disease | 0 | 0
  Cycle 17, Day 28 No Response: number analyzed (Participants) | 1 | 1
  Cycle 17, Day 28 No Response | 0 | 100
  Cycle 20, Day 28 Complete Response: number analyzed (Participants) | 0 | 1
  Cycle 20, Day 28 Complete Response |  | 0
  Cycle 20, Day 28 Partial Response: number analyzed (Participants) | 0 | 1
  Cycle 20, Day 28 Partial Response |  | 0
  Cycle 20, Day 28 Progressive Disease: number analyzed (Participants) | 0 | 1
  Cycle 20, Day 28 Progressive Disease |  | 0
  Cycle 20, Day 28 No Response: number analyzed (Participants) | 0 | 1
  Cycle 20, Day 28 No Response |  | 100
  Final (28 Days post-last dose) Complete Response: number analyzed (Participants) | 4 | 1
  Final (28 Days post-last dose) Complete Response | 50.0 | 0
  Final (28 Days post-last dose) Partial Response: number analyzed (Participants) | 4 | 1
  Final (28 Days post-last dose) Partial Response | 25.0 | 0
  Final (28 Days post-last dose) Progressive Disease: number analyzed (Participants) | 4 | 1
  Final (28 Days post-last dose) Progressive Disease | 0.0 | 0
  Final (28 Days post-last dose) No Response: number analyzed (Participants) | 4 | 1
  Final (28 Days post-last dose) No Response | 25.0 | 100

10. Secondary Outcome: Percentage of All Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants (Irrespective of Spleen Size) by Response Per Modified ELN Criteria
Description: as for outcome 8
Time Frame: Baseline, Day 28 of Cycles 3, 5, 8, 11, 12, 14, 17, 20 and Final visit (28 days after post-last dose)
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Groups:
- All Ruxolitinib-Naïve Participants; All Ruxolitinib-Resistant or Intolerant Participants: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | All Ruxolitinib-Naïve Participants | All Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Percentage of Participants
  Baseline Complete Response | 0 | 0
  Baseline Partial Response | 0 | 0
  Baseline Progressive Disease | 0 | 0
  Baseline No Response | 0 | 0
  Cycle 3, Day 28 Complete Response: number analyzed (Participants) | 19 | 7
  Cycle 3, Day 28 Complete Response | 10.5 | 28.6
  Cycle 3, Day 28 Partial Response: number analyzed (Participants) | 19 | 7
  Cycle 3, Day 28 Partial Response | 68.4 | 42.9
  Cycle 3, Day 28 Progressive Disease: number analyzed (Participants) | 19 | 7
  Cycle 3, Day 28 Progressive Disease | 0 | 0
  Cycle 3, Day 28 No Response: number analyzed (Participants) | 19 | 7
  Cycle 3, Day 28 No Response | 21.1 | 28.6
  Cycle 5, Day 28 Complete Response: number analyzed (Participants) | 16 | 6
  Cycle 5, Day 28 Complete Response | 12.5 | 0
  Cycle 5, Day 28 Partial Response: number analyzed (Participants) | 16 | 6
  Cycle 5, Day 28 Partial Response | 68.8 | 66.7
  Cycle 5, Day 28 Progressive Disease: number analyzed (Participants) | 16 | 6
  Cycle 5, Day 28 Progressive Disease | 0 | 0
  Cycle 5, Day 28 No Response: number analyzed (Participants) | 16 | 6
  Cycle 5, Day 28 No Response | 18.8 | 33.3
  Cycle 8, Day 28 (Week 32) Complete Response: number analyzed (Participants) | 11 | 5
  Cycle 8, Day 28 (Week 32) Complete Response | 18.2 | 20.0
  Cycle 8, Day 28 (Week 32) Partial Response: number analyzed (Participants) | 11 | 5
  Cycle 8, Day 28 (Week 32) Partial Response | 54.5 | 40.0
  Cycle 8, Day 28 (Week 32) Progressive Disease: number analyzed (Participants) | 11 | 5
  Cycle 8, Day 28 (Week 32) Progressive Disease | 0 | 0
  Cycle 8, Day 28 (Week 32) No Response: number analyzed (Participants) | 11 | 5
  Cycle 8, Day 28 (Week 32) No Response | 27.3 | 40.0
  Cycle 11 Day 28 Complete Response: number analyzed (Participants) | 6 | 2
  Cycle 11 Day 28 Complete Response | 16.7 | 0
  Cycle 11 Day 28 Partial Response: number analyzed (Participants) | 6 | 2
  Cycle 11 Day 28 Partial Response | 66.7 | 50.0
  Cycle 11 Day 28 Progressive Disease: number analyzed (Participants) | 6 | 2
  Cycle 11 Day 28 Progressive Disease | 0 | 0
  Cycle 11 Day 28 No Response: number analyzed (Participants) | 6 | 2
  Cycle 11 Day 28 No Response | 16.7 | 50.0
  Cycle 12 Day 28 Complete Response: number analyzed (Participants) | 0 | 1
  Cycle 12 Day 28 Complete Response |  | 0
  Cycle 12 Day 28 Partial Response: number analyzed (Participants) | 0 | 1
  Cycle 12 Day 28 Partial Response |  | 100
  Cycle 12 Day 28 Progressive Disease: number analyzed (Participants) | 0 | 1
  Cycle 12 Day 28 Progressive Disease |  | 0
  Cycle 12 Day 28 No Response: number analyzed (Participants) | 0 | 1
  Cycle 12 Day 28 No Response |  | 0
  Cycle 14, Day 28 Complete Response: number analyzed (Participants) | 6 | 2
  Cycle 14, Day 28 Complete Response | 16.7 | 0
  Cycle 14, Day 28 Partial Response: number analyzed (Participants) | 6 | 2
  Cycle 14, Day 28 Partial Response | 66.7 | 50
  Cycle 14, Day 28 Progressive Disease: number analyzed (Participants) | 6 | 2
  Cycle 14, Day 28 Progressive Disease | 0 | 0
  Cycle 14, Day 28 No Response: number analyzed (Participants) | 6 | 2
  Cycle 14, Day 28 No Response | 16.7 | 50.0
  Cycle 17, Day 28 Complete Response: number analyzed (Participants) | 4 | 2
  Cycle 17, Day 28 Complete Response | 25.0 | 0
  Cycle 17, Day 28 Partial Response: number analyzed (Participants) | 4 | 2
  Cycle 17, Day 28 Partial Response | 25.0 | 0
  Cycle 17, Day 28 Progressive Disease: number analyzed (Participants) | 4 | 2
  Cycle 17, Day 28 Progressive Disease | 0 | 0
  Cycle 17, Day 28 No Response: number analyzed (Participants) | 4 | 2
  Cycle 17, Day 28 No Response | 50.0 | 100
  Cycle 20, Day 28 Complete Response: number analyzed (Participants) | 1 | 1
  Cycle 20, Day 28 Complete Response | 0 | 0
  Cycle 20, Day 28 Partial Response: number analyzed (Participants) | 1 | 1
  Cycle 20, Day 28 Partial Response | 100 | 0
  Cycle 20, Day 28 Progressive Disease: number analyzed (Participants) | 1 | 1
  Cycle 20, Day 28 Progressive Disease | 0 | 0
  Cycle 20, Day 28 No Response: number analyzed (Participants) | 1 | 1
  Cycle 20, Day 28 No Response | 0 | 100
  Final Visit Complete Response: number analyzed (Participants) | 14 | 4
  Final Visit Complete Response | 14.3 | 0
  Final Visit Partial Response: number analyzed (Participants) | 14 | 4
  Final Visit Partial Response | 21.4 | 25.0
  Final Visit Progressive Disease: number analyzed (Participants) | 14 | 4
  Final Visit Progressive Disease | 0 | 0
  Final Visit No Response: number analyzed (Participants) | 14 | 4
  Final Visit No Response | 64.3 | 75.0

11. Secondary Outcome: Percentage of Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly at Baseline With Durable Response Lasting at Least 12 Weeks From Week 32
Description: The percentage of participants with a durable response lasting at least 12 weeks from Week 32 are analyzed by the type of response achieved: Hct control, complete hematologic response, ELN 2009 response criteria, and composite response, if applicable.
  Reported result data start from Cycle 11 Day 28 which is 12 weeks after Week 32 (Cycle 8 Day 28). There was one timepoint for which the participants qualify. The study was pre-maturely terminated by the sponsor decision, therefore did not reach the end of study.
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 Weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly
Number analyzed (Participants) | 15 | 6
Percentage of Participants
  HCT Control: number analyzed (Participants) | 7 | 3
  HCT Control | 42.9 | 100
  Composite Response: number analyzed (Participants) | 7 | 3
  Composite Response | 0 | 0
  ELN Response: number analyzed (Participants) | 8 | 4
  ELN Response | 50 | 75
  Complete Hematologic Response: number analyzed (Participants) | 7 | 3
  Complete Hematologic Response | 28.6 | 66.7

12. Secondary Outcome: Number of Participants With a Durable Response, in Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly at Baseline With Durable Response Lasting at Least 12 Weeks From Week 32
Description: The number of participants with a durable response lasting at least 12 weeks from Week 32 is analyzed by the type of response achieved: Hct control, complete hematologic response, ELN 2009 response criteria, and composite response, if applicable.
  Reported result data start from Cycle 11 Day 28 which is 12 weeks after Week 32 (Cycle 8 Day 28). There was one timepoint for which the participants qualify.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the planned end of study.
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly
Number analyzed (Participants) | 15 | 6
Participants
  HCT Control: number analyzed (Participants) | 7 | 3
  HCT Control | 3 | 3
  Composite Response: number analyzed (Participants) | 7 | 3
  Composite Response | 0 | 0
  ELN Response: number analyzed (Participants) | 8 | 4
  ELN Response | 4 | 3
  Complete Hematologic Response: number analyzed (Participants) | 7 | 3
  Complete Hematologic Response | 2 | 2

13. Secondary Outcome: Percentage of Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly at Baseline With Durable Response Lasting at Least 12 Weeks From Week 32
Description: The percentage of participants with a durable response lasting at least 12 weeks from Week 32 is analyzed by the type of response achieved: Hct control, complete hematologic response, ELN 2009 response criteria, and composite response, if applicable.
  Reported result data start from Cycle 11 Day 28 which is 12 weeks after Week 32 (Cycle 8 Day 28). There was one timepoint for which the participants qualify. The study was pre-maturely terminated by the sponsor decision, therefore did not reach the end of study.
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 Weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 5 | 1
Percentage of Participants
  HCT Control: number analyzed (Participants) | 2 | 1
  HCT Control | 100 | 0
  Composite Response: number analyzed (Participants) | 2 | 1
  Composite Response | 0 | 0
  ELN Response: number analyzed (Participants) | 2 | 1
  ELN Response | 100 | 0
  Complete Hematologic Response: number analyzed (Participants) | 2 | 1
  Complete Hematologic Response | 100 | 0

14. Secondary Outcome: Number of Participants With a Durable Response, in Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly at Baseline With Durable Response Lasting at Least 12 Weeks From Week 32
Description: as for outcome 12
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 5 | 1
Participants
  HCT Control: number analyzed (Participants) | 2 | 1
  HCT Control | 2 | 0
  Composite Response: number analyzed (Participants) | 2 | 1
  Composite Response | 0 | 0
  ELN Response: number analyzed (Participants) | 2 | 1
  ELN Response | 2 | 0
  Complete Hematologic Response: number analyzed (Participants) | 2 | 1
  Complete Hematologic Response | 2 | 0

15. Secondary Outcome: Percentage of All Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants (Irrespective of Spleen Size) With Durable Response Lasting at Least 12 Weeks From Week 32
Description: as for outcome 13
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 Weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Ruxolitinib-Naïve Participants | All Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Percentage of Participants
  After 12 Weeks from Week 32 HCT Control: number analyzed (Participants) | 9 | 4
  After 12 Weeks from Week 32 HCT Control | 55.6 | 75
  After 12 Weeks from Week 32 Composite Response: number analyzed (Participants) | 9 | 4
  After 12 Weeks from Week 32 Composite Response | 0 | 0
  After 12 Weeks from Week 32 ELN Response: number analyzed (Participants) | 10 | 5
  After 12 Weeks from Week 32 ELN Response | 60 | 60
  After 12 Weeks from Week 32 Complete Hematologic Response: number analyzed (Participants) | 9 | 4
  After 12 Weeks from Week 32 Complete Hematologic Response | 44.4 | 50

16. Secondary Outcome: Number of Participants With a Duration Response, in All Ruxolitinib-Naïve and Ruxolitinib-Resistant or Intolerant Participants (Irrespective of Spleen Size) With Durable Response Lasting at Least 12 Weeks From Week 32
Description: as for outcome 12
Time Frame: From Week 32 (Cycle 8 Day 28) and at least 12 weeks after until end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | All Ruxolitinib-Naïve Participants | All Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Participants
  HCT Control: number analyzed (Participants) | 9 | 4
  HCT Control | 5 | 3
  Composite Response: number analyzed (Participants) | 9 | 4
  Composite Response | 0 | 0
  ELN Response: number analyzed (Participants) | 10 | 5
  ELN Response | 6 | 3
  Complete Hematologic Response: number analyzed (Participants) | 9 | 4
  Complete Hematologic Response | 4 | 2

17. Secondary Outcome: Total Number of Participants With Adverse Events by Severity, Graded According to NCI CTCAE v4.0
Description: An adverse event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug. The adverse event severity grading scale for the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v4.0) will be used for assessing adverse event severity.
  During the final analyses, the focus was on the Adverse Events of severity grades >/=3 as shown below. The extensive listings of all grade AEs are available at request.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the planned end of study.
Time Frame: Baseline to end of study (up to 2 years)
Population: ITT population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Participants
  Baseline | 0 | 0 | 0 | 0
  Grade 3-5 AE | 5 | 2 | 3 | 0

18. Secondary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities: Hematology Parameters.
Description: Hematology parameter laboratory values falling outside the standard reference range were planned to be recorded as either high or low.
  There was no clinical laboratory abnormalities identified. The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the end of study.
Time Frame: Baseline to end of study (up to 2 years)
Population: Safety-Evaluable Patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Percentage of Participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities: Clinical Chemistry Parameters
Description: Clinical chemistry parameter laboratory values falling outside the standard reference range were to be recorded as either high or low.
  There was no clinical chemistry abnormalities identified. The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the end of study.
Time Frame: Baseline to end of study (up to 2 years)
Population: Safety-Evaluable Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-Naïve Participants With Splenomegaly | Ruxolitinib-Naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Percentage of Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities: Urinalysis Parameters
Description: Urinalysis parameter laboratory values falling outside the standard reference range were planned to be recorded as either high or low.
  There was no clinical laboratory (urinalysis) abnormalities identified. The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the end of study.
Time Frame: Baseline to end of study (up to 2 years)
Population: ITT population
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Percentage of Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters: PQ(PR), QRS, QT, QTcB, QTcF, and RR Durations
Description: Single 12-lead ECGs was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the planned end of study.
Time Frame: Baseline, Cycle 1 (Day 1, hours 4 and 6, Day 2 pre-dose and 24 Hour, Day 5 pre-dose, 4 and 6 Hour), Cycle 2 (Day 1 pre-dose only), Cycle 3 (Day 1 pre-dose, 4 and 6 Hour), Cycle 4 (Day 1 pre-dose and 4 Hour)
Population: Safety-Evaluable population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Millisecond (msec)
  PR Duration Baseline | 158.93 (24.86) | 153.60 (22.55) | 152.00 (17.39) | 196.00 (0)
  PQ(PR) Durations Cycle 1, Day 1, 4 hour | 0.60 (10.89) | -2.60 (5.37) | -2.00 (9.72) | 4.00 (0)
  PQ(PR) Durations Cycle 1, Day 1, 6 hour | -2.80 (8.10) | -4.40 (15.52) | 6.00 (25.49) | 0.00 (0)
  PQ(PR) Durations Cycle 1, Day 2, pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  PQ(PR) Durations Cycle 1, Day 2, pre-dose | -14.00 (0) | -6.00 (0) |  |
  PQ(PR) Durations Cycle 1, Day 2, 24 hour: number analyzed (Participants) | 14 | 4 | 6 | 1
  PQ(PR) Durations Cycle 1, Day 2, 24 hour | 1.93 (10.32) | 1.00 (16.45) | 0.67 (22.01) | -12.00 (0)
  PQ(PR) Durations Cycle ,1 Day 5, pre-dose: number analyzed (Participants) | 15 | 4 | 5 | 1
  PQ(PR) Durations Cycle ,1 Day 5, pre-dose | -1.00 (11.70) | -12.00 (9.38) | 0.40 (26.59) | -4.00 (0)
  PQ(PR) Durations Cycle 1, Day 5, 4 hour: number analyzed (Participants) | 13 | 4 | 5 | 1
  PQ(PR) Durations Cycle 1, Day 5, 4 hour | -8.00 (12.68) | -6.25 (15.59) | -1.20 (29.52) | 0 (0)
  PQ(PR) Durations Cycle 1, Day 5, 6 hour: number analyzed (Participants) | 13 | 4 | 5 | 1
  PQ(PR) Durations Cycle 1, Day 5, 6 hour | -4.77 (14.08) | -2.75 (10.81) | 7.60 (27.29) | 0 (0)
  PQ(PR) Durations Cycle 2, Day1, pre-dose: number analyzed (Participants) | 14 | 4 | 6 | 1
  PQ(PR) Durations Cycle 2, Day1, pre-dose | 1.43 (14.26) | -5.75 (11.79) | -2.33 (11.89) | -8.00 (0)
  PQ(PR) Durations Cycle 3, Day 1, pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  PQ(PR) Durations Cycle 3, Day 1, pre-dose | -6.00 (0) |  |  |
  PQ(PR) Durations Cycle 3, Day 1, 4 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  PQ(PR) Durations Cycle 3, Day 1, 4 hour | -8.00 (0) |  |  |
  PQ(PR) Durations Cycle 3, Day 1, 6 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  PQ(PR) Durations Cycle 3, Day 1, 6 hour | -6.00 (0) |  |  |
  PQ(PR) Durations Cycle 4, Day 1, pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  PQ(PR) Durations Cycle 4, Day 1, pre-dose | -20.00 (0) |  |  |
  PQ(PR) Durations Cycle 4, Day 1, 4 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  PQ(PR) Durations Cycle 4, Day 1, 4 hour | -20.00 (0) |  |  |
  QRS Duration Baseline | 90.87 (8.25) | 83.80 (6.42) | 83.33 (9.77) | 94.00 (0)
  QRS Cycle 1 Day 1 (4 H) | -1.47 (5.83) | 4.60 (6.69) | 1.33 (1.03) | 0 (0)
  QRS Cycle 1 Day 1 (6 H) | -1.27 (5.27) | 4.00 (3.08) | 0.33 (5.28) | -2.00 (0)
  QRS Cycle 1 Day 2 (PREDOSE): number analyzed (Participants) | 1 | 1 | 0 | 0
  QRS Cycle 1 Day 2 (PREDOSE) | -4.00 (0) | 2.00 (0) |  |
  QRS Cycle 1 Day 2 (24 H): number analyzed (Participants) | 14 | 4 | 6 | 1
  QRS Cycle 1 Day 2 (24 H) | 1.07 (3.77) | 1.75 (6.55) | 3.00 (11.64) | -2.00 (0)
  QRS Cycle 1 Day 5 (PREDOSE): number analyzed (Participants) | 15 | 4 | 5 | 1
  QRS Cycle 1 Day 5 (PREDOSE) | 0.13 (4.63) | 4.00 (9.09) | 0.00 (2.00) | 2.00 (0)
  QRS Cycle 1 Day 5 (4 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QRS Cycle 1 Day 5 (4 H) | -1.08 (3.12) | 3.75 (9.46) | -0.40 (2.61) | 0 (0)
  QRS Cycle 1 Day 5 (6 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QRS Cycle 1 Day 5 (6 H) | -0.92 (4.73) | -0.25 (5.19) | 2.00 (5.83) | 0 (0)
  QRS Cycle 2 Day 1 (PREDOSE): number analyzed (Participants) | 14 | 4 | 6 | 1
  QRS Cycle 2 Day 1 (PREDOSE) | 0.64 (6.25) | 7.75 (9.46) | 1.00 (2.76) | -4.00 (0)
  QRS Cycle 3 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QRS Cycle 3 Day 1 (PREDOSE) | -4.00 (0) |  |  |
  QRS Cycle 3 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QRS Cycle 3 Day 1 (4 H) | -4.00 (0) |  |  |
  QRS Cycle 3 Day 1 (6 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QRS Cycle 3 Day 1 (6 H) | -4.00 (0) |  |  |
  QRS Cycle 4 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QRS Cycle 4 Day 1 (PREDOSE) | -2.00 (0) |  |  |
  QRS Cycle 4 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QRS Cycle 4 Day 1 (4 H) | -2.00 (0) |  |  |
  QT Duration Baseline | 396.67 (31.96) | 392.60 (38.74) | 386.00 (16.78) | 392.00 (0)
  QT Duration Cycle 1 Day 1 (4 H) | -7.33 (26.43) | 16.80 (13.44) | 5.67 (10.07) | 36.00 (0)
  QT Duration Cycle 1 Day 1 (6 H) | -9.40 (23.70) | 11.00 (29.14) | -1.33 (13.49) | 36.00 (0)
  QT Duration Cycle 1 Day 2 (PREDOSE): number analyzed (Participants) | 1 | 1 | 0 | 0
  QT Duration Cycle 1 Day 2 (PREDOSE) | -6.00 (0) | -18.00 (0) |  |
  QT Duration Cycle 1 Day 2 (24 H): number analyzed (Participants) | 14 | 4 | 6 | 1
  QT Duration Cycle 1 Day 2 (24 H) | -10.21 (25.57) | 2.75 (29.00) | 7.00 (16.58) | 0 (0)
  QT Duration Cycle 1 Day 5 (PREDOSE): number analyzed (Participants) | 15 | 4 | 5 | 1
  QT Duration Cycle 1 Day 5 (PREDOSE) | -6.20 (19.79) | -8.75 (21.00) | 8.00 (19.54) | 4.00 (0)
  QT Duration Cycle 1 Day 5 (4 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QT Duration Cycle 1 Day 5 (4 H) | -4.31 (33.31) | 15.25 (15.65) | 3.20 (24.23) | -12.00 (0)
  QT Duration Cycle 1 Day 5 (6 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QT Duration Cycle 1 Day 5 (6 H) | -10.31 (24.83) | 4.75 (20.93) | 7.60 (16.40) | -4.00 (0)
  QT Duration Cycle 2 Day 1 (PREDOSE): number analyzed (Participants) | 14 | 4 | 6 | 1
  QT Duration Cycle 2 Day 1 (PREDOSE) | 5.00 (22.68) | 10.50 (25.96) | 19.00 (13.67) | 12.00 (0)
  QT Durations Cycle 3 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QT Durations Cycle 3 Day 1 (PREDOSE) | -2.00 (0) |  |  |
  QT Durations Cycle 3 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QT Durations Cycle 3 Day 1 (4 H) | -10.00 (0) |  |  |
  QT Durations Cycle 3 Day 1 (6 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QT Durations Cycle 3 Day 1 (6 H) | -4.00 (0) |  |  |
  QT Durations Cycle 4 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QT Durations Cycle 4 Day 1 (PREDOSE) | -16.00 (0) |  |  |
  QT Durations Cycle 4 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QT Durations Cycle 4 Day 1 (4 H) | -16.00 (0) |  |  |
  QTcB baseline | 427.67 (24.23) | 419.60 (7.70) | 424.50 (25.74) | 444.00 (0)
  QTcB - Bazett's Correction Formula Cycle 1 Day 1 (4 H) | 3.80 (12.82) | 21.00 (11.14) | 13.83 (14.05) | -30.00 (0)
  QTcB - Bazett's Correction Formula Cycle 1 Day 1 (6 H) | 8.00 (10.54) | 8.40 (22.40) | 6.33 (5.50) | 5.00 (0)
  QTcB - Bazett's Correction Formula Cycle 1 Day 2 (PREDOSE): number analyzed (Participants) | 1 | 1 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 1 Day 2 (PREDOSE) | -15.00 (0) | -410.00 (0) |  |
  QTcB - Bazett's Correction Formula Cycle 1 Day 2 (24 H): number analyzed (Participants) | 14 | 4 | 6 | 1
  QTcB - Bazett's Correction Formula Cycle 1 Day 2 (24 H) | 3.71 (15.59) | -0.75 (16.40) | 4.50 (14.47) | -14.00 (0)
  QTcB - Bazett's Correction Formula Cycle 1 Day 5 (PREDOSE): number analyzed (Participants) | 15 | 4 | 5 | 1
  QTcB - Bazett's Correction Formula Cycle 1 Day 5 (PREDOSE) | -11.07 (15.21) | -10.00 (8.76) | -9.20 (15.25) | -7.00 (0)
  QTcB - Bazett's Correction Formula Cycle 4 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 4 Day 1 (4 H) | -62.00 (0) |  |  |
  QTcB - Bazett's Correction FormulaCycle 1 Day 5 (4 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QTcB - Bazett's Correction FormulaCycle 1 Day 5 (4 H) | -2.92 (14.20) | 1.50 (8.81) | -4.60 (18.70) | 0.00 (0)
  QTcB - Bazett's Correction Formula Cycle 1 Day 5 (6 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QTcB - Bazett's Correction Formula Cycle 1 Day 5 (6 H) | -4.54 (16.10) | -4.75 (6.18) | -1.60 (15.44) | -12.00 (0)
  QTcB - Bazett's Correction Formula Cycle 2 Day 1 (PREDOSE): number analyzed (Participants) | 14 | 4 | 6 | 1
  QTcB - Bazett's Correction Formula Cycle 2 Day 1 (PREDOSE) | 3.93 (14.42) | 7.75 (20.61) | 0.17 (14.54) | -23.00 (0)
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (PREDOSE) | -16.00 (0) |  |  |
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (4 H) | 6.00 (0) |  |  |
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (6 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 3 Day 1 (6 H) | 8.00 (0) |  |  |
  QTcB - Bazett's Correction Formula Cycle 4 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 4 Day 1 (PREDOSE) | -62.00 (0) |  |  |
  QTcB - Bazett's Correction Formula Cycle 4 Day 1, 4 H: number analyzed (Participants) | 15 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula Cycle 4 Day 1, 4 H | -62.00 (0) |  |  |
  QTcF Durations Fridericia's Correction Formula Baseline | 417.93 (22.41) | 410.00 (17.62) | 411.17 (17.90) | 426.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 1 (4 H) | -1.27 (11.86) | 18.80 (10.08) | 11.67 (11.09) | -8.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 1 (6 H) | 1.00 (8.78) | 10.00 (21.64) | 3.50 (7.37) | 16.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 2 (PREDOSE): number analyzed (Participants) | 1 | 1 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 2 (PREDOSE) | -12.00 (0) | -20.00 (0) |  |
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 2 (24 H): number analyzed (Participants) | 14 | 4 | 6 | 1
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 2 (24 H) | -2.36 (13.32) | 0.00 (20.46) | 5.33 (14.81) | -9.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (PREDOSE): number analyzed (Participants) | 15 | 4 | 5 | 1
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (PREDOSE) | -10.47 (14.17) | -9.25 (8.96) | -3.20 (14.60) | -3.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (4 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (4 H) | -0.08 (26.39) | 4.00 (8.98) | -2.00 (17.36) | -4.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (6 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  QTcF Durations Fridericia's Correction Formula Cycle 1 Day 5 (6 H) | -7.85 (13.44) | -2.25 (8.46) | 1.60 (14.10) | 6.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 2 Day 1 (PREDOSE): number analyzed (Participants) | 14 | 4 | 6 | 1
  QTcF Durations Fridericia's Correction Formula Cycle 2 Day 1 (PREDOSE) | 3.36 (10.49) | 8 (20.51) | 6.83 (12.45) | -11.00 (0)
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (PREDOSE) | -11.00 (0) |  |  |
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (4 H) | 0.00 (0) |  |  |
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (6 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 3 Day 1 (6 H) | 4.00 (0) |  |  |
  QTcF Durations Fridericia's Correction Formula Cycle 4 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 4 Day 1 (PREDOSE) | -45.00 (0) |  |  |
  QTcF Durations Fridericia's Correction Formula Cycle 4 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  QTcF Durations Fridericia's Correction Formula Cycle 4 Day 1 (4 H) | -45.00 (0) |  |  |
  RR Duration Baseline | 861.47 (133.95) | 881.00 (151.46) | 835.83 (139.93) | 779.00 (0)
  RR Duration Cycle 1 Day 1 4 H | -38.87 (130.21) | -5.60 (58.23) | -36.50 (66.76) | 292.00 (0)
  RR Duration Cycle 1 Day 1 6 H | -65.67 (117.44) | 14.00 (100.82) | -31.17 (49.04) | 130.00 (0)
  RR Duration Cycle 1 Day 2 (PREDOSE): number analyzed (Participants) | 1 | 1 | 0 | 0
  RR Duration Cycle 1 Day 2 (PREDOSE) | 28.00 (0) | 18.00 (0) |  |
  RR Duration Cycle 1 Day 2 (24 H): number analyzed (Participants) | 14 | 4 | 6 | 1
  RR Duration Cycle 1 Day 2 (24 H) | -51.50 (121.75) | 17.25 (65.17) | 8.83 (29.78) | 54.00 (0)
  RR Duration Cycle 1 Day 5 (PREDOSE): number analyzed (Participants) | 15 | 4 | 5 | 1
  RR Duration Cycle 1 Day 5 (PREDOSE) | 25.87 (97.32) | -0.75 (104.53) | 67.80 (78.89) | 43.00 (0)
  RR Duration Cycle 1 Day 5 (4 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  RR Duration Cycle 1 Day 5 (4 H) | -26.23 (114.00) | 79.75 (62.99) | 24.20 (114.05) | -47.00 (0)
  RR Duration Cycle 1 Day 5 (6 H): number analyzed (Participants) | 13 | 4 | 5 | 1
  RR Duration Cycle 1 Day 5 (6 H) | -21.46 (121.82) | 49.50 (99.21) | 33.00 (59.05) | -56.00 (0)
  RR Duration Cycle 2 Day 1 (PREDOSE): number analyzed (Participants) | 14 | 4 | 6 | 1
  RR Duration Cycle 2 Day 1 (PREDOSE) | 7.14 (118.26) | 23.75 (86.53) | 78.17 (59.85) | 144.00 (0)
  RR Duration Cycle 3 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  RR Duration Cycle 3 Day 1 (PREDOSE) | 48.00 (0) |  |  |
  RR Duration Cycle 3 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  RR Duration Cycle 3 Day 1 (4 H) | -59.00 (0) |  |  |
  RR Duration Cycle 3 Day 1 (6 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  RR Duration Cycle 3 Day 1 (6 H) | -43.00 (0) |  |  |
  RR Duration Cycle 4 Day 1 (PREDOSE): number analyzed (Participants) | 1 | 0 | 0 | 0
  RR Duration Cycle 4 Day 1 (PREDOSE) | 182.00 (0) |  |  |
  RR Duration Cycle 4 Day 1 (4 H): number analyzed (Participants) | 1 | 0 | 0 | 0
  RR Duration Cycle 4 Day 1 (4 H) | 182.00 (0) |  |  |

22. Secondary Outcome: Change From Baseline in Heart Rate, as Measured by Electrocardiogram
Description: as for outcome 21
Time Frame: as for outcome 21
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Beats per Minute
  Baseline | 71.47 (12.74) | 69.80 (12.28) | 73.17 (10.07) | 77.00 (0)
  Cycle 1, Day 1, 4 Hour | 4.40 (10.58) | 0.60 (5.32) | 2.50 (4.23) | -21.00 (0)
  Cycle 1, Day 1, 6 Hour | 6.20 (10.35) | -0.60 (8.65) | 3.00 (5.44) | -11.00 (0)
  Cycle 1 Day 2, pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Cycle 1 Day 2, pre-dose | -3.00 (0) | -1.00 (0) |  |
  Cycle 1 Day 2, 24 Hour: number analyzed (Participants) | 1 | 4 | 6 | 1
  Cycle 1 Day 2, 24 Hour | 4.71 (10.31) | -1.75 (5.32) | -0.67 (2.50) | -5.00 (0)
  Cycle 1 Day 5, pre-dose: number analyzed (Participants) | 15 | 4 | 5 | 1
  Cycle 1 Day 5, pre-dose | -1.47 (6.56) | -0.75 (8.14) | -5.60 (5.27) | -4.00 (0)
  Cycle 1 Day 5, 4 hour: number analyzed (Participants) | 13 | 4 | 5 | 1
  Cycle 1 Day 5, 4 hour | 2.69 (8.61) | -5.00 (2.94) | -2.20 (7.92) | 5.00 (0)
  Cycle 1 Day 5, 6 hour: number analyzed (Participants) | 13 | 4 | 5 | 1
  Cycle 1 Day 5, 6 hour | 2.23 (9.39) | -3.75 (7.76) | -2.80 (4.92) | 6.00 (0)
  Cycle 2, Day 1, pre-dose: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2, Day 1, pre-dose | -1.43 (9.83) | -1.50 (8.39) | -6.17 (5.19) | -12.00 (0)
  Cycle 3 Day 1, pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1, pre-dose | -5.00 (0) |  |  |
  Cycle 3 Day 1, 4 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1, 4 hour | 7.00 (0) |  |  |
  Cycle 3 Day 1, 6 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1, 6 hour | 5.00 (0) |  |  |
  Cycle 4 Day 1, pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 4 Day 1, pre-dose | -16.00 (0) |  |  |
  Cycle 4 Day 1, 4 hour: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 4 Day 1, 4 hour | -16.00 (0) |  |  |

23. Secondary Outcome: Change From Baseline in Oral Temperature
Description: Vital signs were measured prior to the infusion while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the end of study.
Time Frame: Baseline, Cycle 1 (Days 15 and 22), Cycle 2 and 3 (Days 1 and 15), Each Cycle 4-23 (Day 1 only) and Final Visit
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Degrees Celsius (C)
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Degrees Celsius (C)
  Baseline | 36.50 (0.37) | 36.40 (0.25) | 36.47 (0.28) | 37.10 (0)
  Cycle 1 Day 15 | 0.13 (0.33) | 0.42 (0.50) | 0.18 (0.32) | -0.30 (0)
  Cycle 1 Day 22 | 0.03 (0.18) | 0.04 (0.29) | 0.15 (0.21) | -0.50 (0)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 2 Day 1 | -0.05 (0.28) | 0.05 (0.30) | 0.17 (0.34) | -0.60 (0)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2 Day 15 | 0.04 (0.27) | 0.18 (0.24) | 0.23 (0.38) | -0.30 (0)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 3 Day 1 | -0.09 (0.36) | 0.13 (0.45) | 0.17 (0.43) | 0.10 (0)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 3 | 6 | 1
  Cycle 3 Day 15 | -0.04 (0.31) | -0.03 (0.06) | 0.10 (0.26) | -0.20 (0)
  Cycle 4 Day 1: number analyzed (Participants) | 15 | 3 | 5 | 1
  Cycle 4 Day 1 | -0.05 (0.26) | -0.17 (0.15) | 0.06 (0.37) | -0.50 (0)
  Cycle 5 Day 1: number analyzed (Participants) | 14 | 3 | 5 | 1
  Cycle 5 Day 1 | 0.05 (0.16) | -0.10 (0.36) | 0.10 (0.32) | -0.80 (0)
  Cycle 6 Day 1: number analyzed (Participants) | 12 | 4 | 5 | 1
  Cycle 6 Day 1 | -0.03 (0.16) | -0.10 (0.45) | 0.12 (0.16) | -0.40 (0)
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 2 | 3 | 1
  Cycle 7 Day 1 | 0.01 (0.30) | -0.20 (0.28) | 0.20 (0.26) | -0.60 (0)
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 2 | 4 | 1
  Cycle 8 Day 1 | -0.01 (0.20) | -0.05 (0.64) | 0.20 (0.36) | -0.30 (0)
  Cycle 9 Day 1: number analyzed (Participants) | 7 | 2 | 3 | 1
  Cycle 9 Day 1 | 0.03 (0.13) | 0.05 (0.35) | -0.07 (0.42) | -0.40 (0)
  Cycle 10 Day 1: number analyzed (Participants) | 6 | 2 | 3 | 1
  Cycle 10 Day 1 | -0.08 (0.10) | 0.30 (0.42) | 0.10 (0.35) | -0.60 (0)
  Cycle 11 Day 1: number analyzed (Participants) | 6 | 1 | 2 | 1
  Cycle 11 Day 1 | -0.07 (0.19) | -0.20 (0) | -0.10 (0.14) | -0.40 (0)
  Cycle 12 Day 1: number analyzed (Participants) | 5 | 1 | 2 | 1
  Cycle 12 Day 1 | -0.10 (0.16) | 0.30 (0) | -0.20 (0.14) | -0.70 (0)
  Cycle 13 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 13 Day 1 | 0.00 (0.19) | -0.70 (0) | 0 | -0.70 (0)
  Cycle 14 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 14 Day 1 | 0.00 (0.41) | -0.10 (0) | -0.30 (0) | -0.70 (0)
  Cycle 15 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 15 Day 1 | -0.10 (0.14) | -0.30 (0) | -0.40 (0) | -0.50 (0)
  Cycle 16 Day 1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Cycle 16 Day 1 | 0.03 (0.30) | -0.80 (0) | -0.10 (0) | -0.50 (0)
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 1
  Cycle 17 Day 1 | 0.03 (0.12) | 0.60 (0) | 0.00 (60) | -0.80 (0)
  Cycle 18 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 1
  Cycle 18 Day 1 | 0.07 (0.15) |  | -0.20 (0) | -0.80 (0)
  Cycle 19 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 19 Day 1 | -0.15 (0.21) |  | 0 | -0.50 (0)
  Cycle 20 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 20 Day 1 | 0.00 (0.14) |  | 0 | -0.50 (0)
  Cycle 21 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 21 Day 1 | 0 (0) |  |  | -0.40 (0)
  Cycle 22 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 22 Day 1 | -0.50 (0) |  |  | -0.70 (0)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Cycle 23 Day 1 |  |  |  | -0.80 (0)
  Final Visit: number analyzed (Participants) | 12 | 5 | 5 | 1
  Final Visit | -0.08 (0.15) | 0.26 (0.26) | 0.08 (0.37) | -0.50 (0)

24. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital signs were measured prior to the infusion while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the planned end of study.
Time Frame: Baseline, Cycle 1 (Days 15 and 22), Cycle 2 and 3 (Days 1 and 15), Each Cycle 4-23 (Day 1 only) and Final Visit
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Beats per Minute
  Baseline | 74.7 (12.3) | 71.6 (9.2) | 76.7 (14.1) | 68.0 (0)
  Cycle 1 Day 15 | 4.5 (13.2) | 5.4 (5.5) | -0.7 (4.8) | 7.0 (0)
  Cycle 1 Day 22 | 3.9 (11.3) | 8.2 (4.9) | -5.8 (3.9) | 8.0 (0)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 2 Day 1 | -1.1 (8.6) | 1.8 (8.7) | -9.3 (6.1) | 12.0 (0)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2 Day 15 | 0.1 (11.0) | 1.8 (8.5) | -5.8 (5.5) | 9.0 (0)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 3 Day 1 | -2.8 (9.4) | -2.0 (8.6) | -4.2 (9.9) | 9.0 (0)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 3 Day 15 | -1.2 (9.7) | 10.8 (13.6) | -2.2 (11.0) | 21.0 (0)
  Cycle 4 Day 1: number analyzed (Participants) | 15 | 3 | 5 | 1
  Cycle 4 Day 1 | 1.0 (11.2) | 1.7 (9.9) | -6.6 (9.8) | 24.0 (0)
  Cycle 5 Day 1: number analyzed (Participants) | 14 | 4 | 5 | 1
  Cycle 5 Day 1 | 0.6 (8.4) | -4.0 (9.3) | -3.6 (4.2) | 28.0 (0)
  Cycle 6 Day 1: number analyzed (Participants) | 12 | 4 | 5 | 1
  Cycle 6 Day 1 | 0.4 (9.1) | -4.3 (6.8) | -1.6 (6.8) | 14.0 (0)
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 2 | 3 | 1
  Cycle 7 Day 1 | 1.4 (14.6) | 1.5 (16.3) | -1.0 (9.8) | 21.0 (0)
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 2 | 4 | 1
  Cycle 8 Day 1 | -3.9 (13.3) | -1.0 (12.7) | 0.5 (3.1) | 11.0 (0)
  Cycle 9 Day 1: number analyzed (Participants) | 7 | 2 | 3 | 1
  Cycle 9 Day 1 | -5.4 (6.4) | 0.0 (5.7) | 0.3 (2.5) | 0 (0)
  Cycle 10 Day 1: number analyzed (Participants) | 6 | 2 | 3 | 1
  Cycle 10 Day 1 | -0.3 (9.9) | 8.5 (19.1) | 2.3 (8.5) | 20.0 (0)
  Cycle 11 Day 1: number analyzed (Participants) | 6 | 1 | 2 | 1
  Cycle 11 Day 1 | -2.5 (11.5) | -2.0 (0) | 2.5 (0.7) | 37.0 (0)
  Cycle 12, Day 1: number analyzed (Participants) | 5 | 1 | 2 | 1
  Cycle 12, Day 1 | -0.2 (11.6) | -6.0 (0) | -1.0 (4.2) | 21.0 (0)
  Cycle 13, Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 13, Day 1 | -2.8 (7.8) | -5.0 (0) | -1.0 (0) | 16.0 (0)
  Cycle 14, Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 14, Day 1 | -3.8 (11.1) | -2.0 (0) | -4.0 (0) | 12.0 (0)
  Cycle 15 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 15 Day 1 | -0.8 (10.4) | 10.0 (0) | -2.0 (0) | 14.0 (0)
  Cycle 16 Day 1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Cycle 16 Day 1 | -1.3 (15.6) | -2.0 (0) | -2.0 (0) | 16.0 (0)
  Cycle 17, Day 1: number analyzed (Participants) | 3 | 1 | 1 | 1
  Cycle 17, Day 1 | -12.7 (9.5) | 9.0 (0) | 1.0 (0) | 22.0 (0)
  Cycle 18, Day 1: number analyzed (Participants) | 3 | 0 | 1 | 1
  Cycle 18, Day 1 | -4.3 (3.5) |  | -3.0 (0) | 16.0 (0)
  Cycle 19, Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 19, Day 1 | -9.0 (5.7) |  | 6.0 (0) | 15.0 (0)
  Cycle 20, Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 20, Day 1 | -5.0 (9.9) |  | 4.0 (0) | 5.0 (0)
  Cycle 21, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 21, Day 1 | 2.0 (0) |  |  | 17.0 (0)
  Cycle 22, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 22, Day 1 | -8.0 (0) |  |  | 14 (0)
  Cycle 23, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Cycle 23, Day 1 |  |  |  | 19.0 (0)
  Final Visit: number analyzed (Participants) | 12 | 5 | 5 | 1
  Final Visit | -1.7 (12.2) | 0.2 (11.6) | 0.2 (10.1) | 16.0 (0)

25. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: as for outcome 24
Time Frame: Baseline, Cycle 1 (Days 15 and 22), Cycle 2 and 3 (Days 1 and 15), Each Cycle 4-23 (Day 1 only) and Final Visit
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Breaths per Minute
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Breaths per Minute
  Baseline | 17.4 (2.0) | 17.4 (1.9) | 18.2 (2.6) | 16.0 (0)
  Cycle 1 Day 15 | -0.3 (1.0) | -0.2 (1.8) | -0.2 (1.8) | 0 (0)
  Cycle 1 Day 22 | -0.5 (0.8) | 0.2 (0.4) | -0.5 (2.2) | 0 (0)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 4 | 5 | 1
  Cycle 2 Day 1 | -0.3 (1.5) | -0.3 (1.7) | -0.4 (1.7) | 0 (0)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2 Day 15 | -0.2 (1.0) | 0.0 (0.8) | -1.2 (1.8) | 2.0 (0)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 4 | 5 | 1
  Cycle 3 Day 1 | -0.7 (1.3) | -1.5 (3.1) | -1.8 (1.8) | 0 (0)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 3 | 5 | 1
  Cycle 3 Day 15 | -0.7 (1.3) | 0.0 (1.0) | -1.0 (1.0) | 0 (0)
  Cycle 4 Day 1: number analyzed (Participants) | 15 | 3 | 5 | 1
  Cycle 4 Day 1 | -0.3 (1.3) | -3.3 (4.2) | -1.0 (1.0) | 2.0 (0)
  Cycle 5 Day 1: number analyzed (Participants) | 14 | 3 | 5 | 1
  Cycle 5 Day 1 | -0.4 (1.9) | -0.3 (0.6) | 1.0 (2.2) | 0 (0)
  Cycle 6 Day 1: number analyzed (Participants) | 12 | 4 | 5 | 1
  Cycle 6 Day 1 | -0.5 (1.3) | -0.5 (1.9) | -0.6 (1.3) | 2.0 (0)
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 2 | 3 | 1
  Cycle 7 Day 1 | -0.2 (1.7) | 0 (0) | -2.3 (1.5) | 2.0 (0)
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 2 | 4 | 1
  Cycle 8 Day 1 | 0.1 (1.5) | -0.5 (2.1) | -0.8 (3.8) | 0 (0)
  Cycle 9 Day 1: number analyzed (Participants) | 7 | 2 | 3 | 1
  Cycle 9 Day 1 | 0.4 (1.8) | 0.5 (0.7) | -1.7 (6.0) | -2.0 (0)
  Cycle 10 Day 1: number analyzed (Participants) | 6 | 2 | 3 | 1
  Cycle 10 Day 1 | -0.2 (1.6) | -0.5 (2.1) | -0.3 (5.5) | 0 (0)
  Cycle 11 Day 1: number analyzed (Participants) | 6 | 1 | 2 | 1
  Cycle 11 Day 1 | -0.8 (1.0) | 1.0 (0) | -0.5 (0.7) | 2.0 (0)
  Cycle 12 Day 1: number analyzed (Participants) | 5 | 1 | 2 | 1
  Cycle 12 Day 1 | -0.4 (1.5) | 1.0 (0) | 1.5 (0.7) | 0 (0)
  Cycle 13 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 13 Day 1 | -1.4 (2.8) | 1.0 (0) | -1.0 (0) | 2.0 (0)
  Cycle 14 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 14 Day 1 | 0.8 (2.3) | 1.0 (0) | 1.0 (0) | 0 (0)
  Cycle 15 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 15 Day 1 | 0.0 (1.4) | 1.0 (0) | -1.0 (0) | 0 (0)
  Cycle 16 Day 1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Cycle 16 Day 1 | -0.3 (1.3) | 1.0 (0) | -2.0 (0) | 0 (0)
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 1
  Cycle 17 Day 1 | 1.3 (2.3) | 1.0 (0) | -2.0 (0) | 0 (0)
  Cycle 18 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 1
  Cycle 18 Day 1 | 1.3 (2.3) |  | -1.0 (0) | 2.0 (0)
  Cycle 19 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 19 Day 1 | 1.5 (2.1) |  | -3.0 (0) | 2.0 (0)
  Cycle 20 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 20 Day 1 | 2.0 (2.8) |  | -3.0 (0) | 2.0 (0)
  Cycle 21 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 21 Day 1 | 2.0 (0) |  |  | 0 (0)
  Cycle 22 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 22 Day 1 | 0.0 (0) |  |  | 0 (0)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Cycle 23 Day 1 |  |  |  | 0 (0)
  Final visit: number analyzed (Participants) | 12 | 5 | 5 | 1
  Final visit | -0.3 (1.5) | -1.2 (1.5) | -1.8 (1.8) | 0 (0)

26. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: as for outcome 24
Time Frame: Baseline, Cycle 1 (Days 15 and 22), Cycle 2 and 3 (Days 1 and 15), Each Cycle 4-23 (Day 1 only) and Final Visit
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Millimeters of mercury (mmHg)
  Baseline | 129.3 (11.5) | 132.0 (17.2) | 122.3 (16.9) | 106.0 (0)
  Cycle 1, Day 15 | 4.4 (9.9) | 3.6 (13.6) | 3.8 (15.1) | 5.0 (0)
  Cycle 1, Days 22 | 3.3 (9.4) | -5.6 (11.8) | 4.8 (10.1) | -5.0 (0)
  Cycle 2, Day 1: number analyzed (Participants) | 13 | 4 | 6 | 1
  Cycle 2, Day 1 | 3.0 (10.3) | 2.8 (8.4) | -4.3 (7.9) | 10.0 (0)
  Cycle 2 , Day 15: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2 , Day 15 | 5.2 (9.8) | -2.0 (13.6) | -7.2 (9.6) | 30.0 (0)
  Cycle 3, Day 1: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 3, Day 1 | 5.5 (10.8) | -3.0 (9.8) | 7.3 (18.3) | 0 (0)
  Cycle 3, Day 15: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 3, Day 15 | 1.2 (11.2) | -3.5 (14.2) | -3.8 (16.7) | 6.0 (0)
  Cycle 4, Day 1: number analyzed (Participants) | 15 | 3 | 6 | 1
  Cycle 4, Day 1 | 2.2 (9.1) | -7.3 (9.3) | 9.8 (8.1) | 13.0 (0)
  Cycle 5, Day 1: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 5, Day 1 | 4.2 (10.5) | -2.5 (6.8) | 3.3 (6.9) | 16.0 (0)
  Cycle 6 Day 1: number analyzed (Participants) | 12 | 4 | 5 | 1
  Cycle 6 Day 1 | 11.2 (13.0) | 2.5 (9.7) | 8.6 (10.8) | 8.0 (0)
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 2 | 3 | 1
  Cycle 7 Day 1 | 4.7 (4.2) | -4.0 (15.6) | 10.0 (5.0) | 29.0 (0)
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 2 | 4 | 1
  Cycle 8 Day 1 | 8.8 (9.0) | 5.0 (7.1) | 14.0 (18.8) | 9.0 (0)
  Cycle 9 Day 1: number analyzed (Participants) | 7 | 2 | 3 | 1
  Cycle 9 Day 1 | 12.6 (8.3) | 3.0 (9.9) | -4.3 (4.9) | 26.0 (0)
  Cycle 10 Day 1: number analyzed (Participants) | 6 | 2 | 3 | 1
  Cycle 10 Day 1 | 11.8 (9.9) | -3.0 (2.8) | 11.0 (13.2) | 30.0 (0)
  Cycle 11 Day 1: number analyzed (Participants) | 6 | 1 | 2 | 1
  Cycle 11 Day 1 | 8.5 (12.3) | 14.0 (0) | 11.0 (12.7) | 34.0 (0)
  Cycle 12 Day 1: number analyzed (Participants) | 5 | 1 | 2 | 1
  Cycle 12 Day 1 | 10.8 (11.5) | -8.0 (0) | 6.5 (3.5) | 6.0 (0)
  Cycle 13 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 13 Day 1 | 13.4 (5.1) | -8.0 (0) | 8.0 (0) | 14.0 (0)
  Cycle 14 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 14 Day 1 | 4.4 (14.7) | 18.0 (0) | 3.0 (0) | 14.0 (0)
  Cycle 15 Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 15 Day 1 | 13.6 (7.5) | 14.0 (0) | 4.0 (0) | 5.0 (0)
  Cycle 16 Day 1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Cycle 16 Day 1 | 7.5 (8.6) | 8.0 (0) | 9.0 (0) | 4.0 (0)
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 1
  Cycle 17 Day 1 | 9.3 (5.8) | 24.0 (0) | 7.0 (0) | 6.0 (0)
  Cycle 18 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 1
  Cycle 18 Day 1 | 5.7 (4.2) |  | 9.0 (0) | 13.0 (0)
  Cycle 19 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 19 Day 1 | 2.5 (3.5) |  | 9.0 (0) | 13.0 (0)
  Cycle 20 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 20 Day 1 | 11.5 (9.2) |  | 9.0 (0) | 13.0 (0)
  Cycle 21 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 21 Day 1 | -18.0 (0) |  |  | 7.0 (0)
  Cycle 22 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 22 Day 1 | 24.0 (0) |  |  | 6.0 (0)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Cycle 23 Day 1 |  |  |  | 11.0 (0)
  Final Visit: number analyzed (Participants) | 12 | 5 | 5 | 1
  Final Visit | 1.3 (9.7) | 7.6 (16.2) | 12.8 (23.9) | 19.0 (0)

27. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: as for outcome 24
Time Frame: Baseline, Cycle 1 (Days 15 and 22), Cycle 2 and 3 (Days 1 and 15), Each Cycle 4-23 (Day 1 only) and Final Visit
Population: Safety-Evaluable Participants. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Millimeters of mercury (mmHg)
  Baseline | 76.3 (7.8) | 73.2 (5.2) | 72.3 (9.0) | 65.0 (0)
  Cycle1, Day 15 | 5.1 (8.7) | 10.0 (8.7) | -1.8 (3.4) | 0.0 (0)
  Cycle 1, Day 22 | 3.6 (6.1) | 2.4 (3.2) | -2.2 (5.8) | -1.0 (0)
  Cycle 2, Day 1: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 2, Day 1 | 6.1 (8.3) | 3.0 (2.9) | -0.2 (9.3) | 3.0 (0)
  Cycle 2, Day 15: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 2, Day 15 | 4.1 (6.3) | 2.5 (9.7) | -5.5 (3.4) | 16.0 (0)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 4 | 6 | 1
  Cycle 3 Day 1 | 6.2 (8.1) | 5.8 (10.0) | -4.0 (12.4) | 5.0 (0)
  Cycle 3, Day 15: number analyzed (Participants) | 15 | 4 | 6 | 1
  Cycle 3, Day 15 | 1.8 (10.5) | 2.0 (10.1) | -7.5 (7.0) | 8.0 (0)
  Cycle 4, Day 1: number analyzed (Participants) | 15 | 3 | 5 | 1
  Cycle 4, Day 1 | 5.5 (5.7) | 2.7 (6.8) | -0.4 (5.0) | 1.0 (0)
  Cycle 5, Day 1: number analyzed (Participants) | 14 | 4 | 4 | 1
  Cycle 5, Day 1 | 1.7 (6.1) | 5.0 (5.8) | -5.0 (4.5) | 1.0 (0)
  Cycle 6, Day 1: number analyzed (Participants) | 12 | 4 | 5 | 1
  Cycle 6, Day 1 | 5.9 (4.5) | 3.3 (11.1) | -2.0 (9.5) | 12.0 (0)
  Cycle 7, Day 1: number analyzed (Participants) | 11 | 2 | 3 | 1
  Cycle 7, Day 1 | 2.9 (4.8) | 4.5 (13.4) | -5.3 (9.0) | 30.0 (0)
  Cycle 8, Day 1: number analyzed (Participants) | 9 | 2 | 4 | 1
  Cycle 8, Day 1 | 7.8 (5.4) | 5.0 (7.1) | 0.5 (12.3) | 10.0 (0)
  Cycle 9, Day 1: number analyzed (Participants) | 7 | 2 | 3 | 1
  Cycle 9, Day 1 | 4.1 (8.4) | 4.0 (5.7) | -2.7 (1.5) | 4.0 (0)
  Cycle 10, Day 1: number analyzed (Participants) | 6 | 2 | 3 | 1
  Cycle 10, Day 1 | 3.7 (5.9) | 5.0 (0) | -2.3 (10.1) | 3.0 (0)
  Cycle 11, Day 1: number analyzed (Participants) | 6 | 1 | 2 | 1
  Cycle 11, Day 1 | 9.7 (14.1) | 10.0 (0) | 1.0 (7.1) | 24.0 (0)
  Cycle 12, Day 1: number analyzed (Participants) | 5 | 1 | 2 | 1
  Cycle 12, Day 1 | 9.8 (8.6) | 6.0 (0) | 2.0 (4.2) | 8.0 (0)
  Cycle 13, Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 13, Day 1 | 9.0 (7.6) | 4.0 (0) | 2.0 (0) | 10.0 (0)
  Cycle 14, Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 14, Day 1 | 5.6 (5.1) | 19.0 (0) | -9.0 (0) | 11.0 (0)
  Cycle 15, Day 1: number analyzed (Participants) | 5 | 1 | 1 | 1
  Cycle 15, Day 1 | 7.0 (8.0) | 10.0 (0) | -2.0 (0) | 7.0 (0)
  Cycle 16, Day 1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Cycle 16, Day 1 | 9.8 (7.8) | 11.0 (0) | 7.0 (0) | 6.0 (0)
  Cycle 17, Day 1: number analyzed (Participants) | 3 | 1 | 1 | 1
  Cycle 17, Day 1 | 11.3 (3.5) | 11.0 (0) | 3.0 (0) | 7.0 (0)
  Cycle 18, Day 1: number analyzed (Participants) | 3 | 0 | 1 | 1
  Cycle 18, Day 1 | 5.0 (1.7) |  | -2.0 (0) | 3.0 (0)
  Cycle 19, Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 19, Day 1 | 4.0 (5.7) |  | 5.0 (0) | 8.0 (0)
  Cycle 20, Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 20, Day 1 | 12.5 (3.5) |  | -1.0 (0) | 2.0 (0)
  Cycle 21, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 21, Day 1 | -3.0 (0) |  |  | 7.0 (0)
  Cycle 22, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Cycle 22, Day 1 | 22.0 (0) |  |  | 8.0 (0)
  Cycle 23, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Cycle 23, Day 1 |  |  |  | 7.0 (0)
  Final visit: number analyzed (Participants) | 12 | 5 | 5 | 1
  Final visit | 5.8 (9.0) | 3.8 (14.0) | -2.0 (12.6) | 11.0 (0)

28. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status Over Time
Description: The ECOG performance status is a scale used to quantify cancer patients' general well-being and activities of daily life. The scale ranges from 0 to 5, with 0 denoting perfect health and 5 indicating death. The 6 categories are 0=Asymptomatic (Fully active, able to carry on all pre-disease activities without restriction), 1=Symptomatic but completely ambulatory, 2=Symptomatic, < 50% in bed during the day (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours), 3=Symptomatic, > 50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours), 4=Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair), 5=Death.
  Only baseline data were collectable. The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the planned end of study.
Time Frame: Baseline
Population: Safety-Evaluable Patients. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participant
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Percentage of Participant
  Baseline 0 | 66.7 | 60.0 | 50.0 | 100.0
  Baseline 1 | 33.3 | 40.0 | 50.0 | 0

29. Secondary Outcome: Percentage of Participants With Concomitant Medications
Description: Participants with Concomitant Medications used from 28 days prior to screening until the final visit or end of study (EOS) were reported.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Overall Study Period
Population: Safety-Evaluable Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Groups:
- Ruxolitinib-naïve Participants Without SplenomegalyEdit; Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
- Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly: t Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | Ruxolitinib-naïve Participants With Splenomegaly | Ruxolitinib-naïve Participants Without SplenomegalyEdit | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
Number analyzed (Participants) | 15 | 5 | 6 | 1
Percentage of Participants | 100 | 100 | 100 | 100

30. Secondary Outcome: Maximum Serum Concentration Observed (Cmax) of Idasanutlin
Description: Cmax is the maximum observed concentration of drug in blood. The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine Cmax as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Groups:
- Ruxolitinib-Naïve ParticipantsEditEdit; Ruxolitinib-Resistant or Intolerant Participants: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | Ruxolitinib-Naïve ParticipantsEditEdit | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Trough Concentration (Ctrough) of Idasanutlin
Description: Ctrough is the measured concentration of a drug at the end of a dosing interval at steady state.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine Ctrough as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Groups:
- Ruxolitinib-Naïve Participants; Ruxolitinib-Resistant or Intolerant Participants: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Time of Maximum Concentration Observed (Tmax) of Idasanutlin
Description: Tmax is the time elapsed from the time of drug administration to maximum plasma concentration.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine tmax as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Clearance (CL) of Idasanutlin
Description: CL is a measure of the body's elimination of a drug from plasma over time. The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine CL as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Apparent Clearance (CL/F) of Idasanutlin
Description: CL/F is a measure of the body's elimination of a drug from plasma over time, after oral administration.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine CL/F as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Volume or Apparent Volume of Distribution (Vdss/F) of Idasanutlin
Description: Vdss/F is the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the plasma.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine Vdss/F as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Idasanutlin
Description: AUC (from zero to infinity) represents the total drug exposure over time. The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine AUC as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Half-life (t1/2) of Idasanutlin
Description: t1/2 is defined as the time required for the drug plasma concentration to be reduced to half.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: Days 1, 2, and 5 of Cycles 1 and 4
Population: The study plan was to determine t1/2 as part of the pharmacokinetics, however study was terminated prematurely in the initial phase after 27 patients were recruited due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity leading to high dropout rate in participants. Therefore, no participants were available for this endpoint and result data were not collected.
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Baseline and Mean Change From Baseline Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) Over Time
Description: MPN-SAF Total Symptom Score is the sum of the following 10 items: early satiety, abdominal discomfort, inactivity, concentration issues, night sweats, Itching, Bone pain, Fever and Unintentional weight loss last 6 months and fatigue. The participant provides a severity score for each symptom on a scale of 0 as a minimum score (none/absent) to 10 (worst imaginable) as a maximum score.
  Baseline (Cycle 1, Day 1) MPN-SAF total symptom score and the mean change from baseline score at each timepoint are reported. The change from baseline score was calculated by subtracting the post-baseline score from the baseline score.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the end of study.
Time Frame: Baseline (Cycle 1 Day 1), Cycle 2 Day 1, Days 28 of Cycles 3, 5, 8 (Week 32), 11, 14, 17 ) Day 28, Cycle 5 Day 28, End of Cycle 8 (Week 32), and Final Visit
Population: ITT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Score on a Scale
  Baseline (Cycle 1 Day 1): number analyzed (Participants) | 19 | 6
  Baseline (Cycle 1 Day 1) | 31.95 (19.95) | 26.00 (11.83)
  Cycle 2 Day 1: number analyzed (Participants) | 17 | 5
  Cycle 2 Day 1 | -5.06 (12.91) | 0.80 (26.37)
  Cycle 3 Day 28: number analyzed (Participants) | 16 | 5
  Cycle 3 Day 28 | -6.38 (12.71) | -8.00 (15.08)
  Cycle 5 Day 28,: number analyzed (Participants) | 12 | 6
  Cycle 5 Day 28, | -7.00 (12.72) | -9.50 (10.56)
  Week 32: number analyzed (Participants) | 10 | 5
  Week 32 | -8.20 (12.79) | -5.00 (15.26)
  Cycle 11 Day 28: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 | -4.60 (3.71) | -7.50 (3.54)
  Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 | -4.67 (5.54) | -10.50 (4.95)
  Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 | -3.25 (5.38) | -12.00 (1.41)
  Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 | -12.00 (0) | -8.00 (0)
  Final Visit: number analyzed (Participants) | 13 | 5
  Final Visit | -5.92 (9.96) | -7.20 (5.63)

39. Secondary Outcome: Baseline and Mean Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Scores Over Time
Description: Reported EORTC QLQ-C30 Scores include: Cognitive function, Diarrhea Emotional functioning, Nausea and vomiting, Social functioning, Physical functioning, Global health status/QoL and Role functioning. The questions use a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores are averaged and transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
  The study was pre-maturely terminated by the sponsor's decision due to non-transformative efficacy and poor long-term tolerability of the dosing schedule as well as due to chronic gastrointestinal toxicity, therefore did not reach the end of study.
Time Frame: Baseline (Cycle 1 Day 1), Cycle 2 Day 1, Cycles 3, 5, 8, 11, 14, 17, 20 Day 28 and Final Visit
Population: ITT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Score on a Scale
  EORTC QLQ-C30 Scores: Cognitive function Baseline | 65.83 (32.21) | 76.19 (30.21)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 2, Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Cognitive function Cycle 2, Day 1 | 11.11 (11.43) | 8.33 (13.94)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Cognitive function Cycle 3 Day 28 | 7.02 (16.02) | 6.67 (19.00)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 5 Day 28: number analyzed (Participants) | 14 | 7
  EORTC QLQ-C30 Scores: Cognitive function Cycle 5 Day 28 | 1.19 (22.13) | 11.11 (25.09)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Cognitive function Cycle 8 (Week 32) | 6.06 (18.67) | -3.33 (21.73)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Cognitive function Cycle 11 Day 28 | 8.33 (13.94) | 0 (0)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Cognitive function Cycle 14 Day 28 | 5.56 (17.21) | 0 (0)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Cognitive function Cycle 17 Day 28 | 0.00 (13.61) | -8.33 (11.79)
  EORTC QLQ-C30 Scores: Cognitive function Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Cognitive function Cycle 20 Day 28 | 0 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Cognitive function Final Visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Cognitive function Final Visit | 4.44 (18.33) | 6.67 (9.13)
  EORTC QLQ-C30 Scores: Diarrhea Baseline | 8.33 (18.34) | 14.29 (17.82)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 2 Day 1: number analyzed (Participants) | 18 | 7
  EORTC QLQ-C30 Scores: Diarrhea Cycle 2 Day 1 | -5.56 (17.15) | 5.56 (13.61)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Diarrhea Cycle 3 Day 28 | 1.75 (17.48) | 0 (0)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Diarrhea Cycle 5 Day 28 | 7.14 (19.30) | 5.56 (13.61)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Diarrhea Cycle 8 (Week 32) | 9.09 (26.21) | 20.00 (18.26)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Diarrhea Cycle 11 Day 28 | 5.56 (13.61) | 0 (0)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Diarrhea Cycle 14 Day 28 | 5.56 (13.61) | 0 (0)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Diarrhea Cycle 17 Day 28 | 25.00 (31.91) | 0 (0)
  EORTC QLQ-C30 Scores: Diarrhea Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Diarrhea Cycle 20 Day 28 | 0 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Diarrhea Final visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Diarrhea Final visit | 13.33 (32.85) | 6.67 (14.91)
  EORTC QLQ-C30 Scores: Emotional functioning Baseline | 65.83 (28.34) | 64.29 (21.36)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 1 Day 28: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 1 Day 28 | 13.43 (20.24) | 15.28 (13.35)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 3 Day 28 | 14.04 (21.88) | 8.33 (10.21)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 5 Day 28 | 16.07 (20.53) | 6.94 (16.17)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 8 (Week 32) | 14.39 (18.29) | 5.00 (27.39)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 11 Day 28 | 6.94 (11.08) | 16.67 (0)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 14 Day 28 | 5.56 (10.09) | -4.17 (5.89)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 17 Day 28 | -8.33 (16.67) | 0 (0)
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Emotional functioning Cycle 20 Day 28 | 0 (0) | 8.33 (0)
  EORTC QLQ-C30 Scores: Emotional functioning Final visit: number analyzed (Participants) | 20 | 5
  EORTC QLQ-C30 Scores: Emotional functioning Final visit | 3.33 (18.31) | 16.67 (18.63)
  EORTC QLQ-C30 Scores: Nausea and vomiting Baseline | 10.00 (16.58) | 2.38 (6.30)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 2 Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 2 Day 1 | -4.63 (12.53) | 8.33 (22.97)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 3 Day 28 | -1.75 (17.48) | 3.33 (13.94)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 5 Day 28 | -2.38 (11.05) | 8.33 (17.48)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 8 (Week 32) | 7.58 (23.99) | 16.67 (16.67)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 11 Day 28 | 2.78 (12.55) | 0.00 (23.57)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 14 Day 28 | -2.78 (6.80) | -8.33 (11.79)
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Nausea and vomiting Cycle 20 Day 28 | 0 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Nausea and vomiting Final visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Nausea and vomiting Final visit | 11.11 (33.73) | 6.67 (19.00)
  EORTC QLQ-C30 Scores: Social functioning Baseline | 67.50 (35.24) | 76.19 (13.11)
  EORTC QLQ-C30 Scores: Social functioning Cycle 2 Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Social functioning Cycle 2 Day 1 | 4.63 (12.53) | 0.00 (10.54)
  EORTC QLQ-C30 Scores: Social functioning Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Social functioning Cycle 3 Day 28 | -1.75 (22.15) | 3.33 (13.94)
  EORTC QLQ-C30 Scores: Social functioning Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Social functioning Cycle 5 Day 28 | 5.95 (24.98) | -2.78 (26.70)
  EORTC QLQ-C30 Scores: Social functioning Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Social functioning Cycle 8 (Week 32) | 0.00 (18.26) | -6.67 (19.00)
  EORTC QLQ-C30 Scores: Social functioning Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Social functioning Cycle 11 Day 28 | 0.00 (18.26) | 0 (0)
  EORTC QLQ-C30 Scores: Social functioning Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Social functioning Cycle 14 Day 28 | 0.00 (10.54) | 0 (0)
  EORTC QLQ-C30 Scores: Social functioning Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Social functioning Cycle 17 Day 28 | -4.17 (8.33) | 0 (0)
  EORTC QLQ-C30 Scores: Social functioning Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Social functioning Cycle 20 Day 28 | 0 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Social functioning Final visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Social functioning Final visit | 0.00 (30.86) | -6.67 (25.28)
  EORTC QLQ-C30 Scores: Physical functioning Baseline | 86.33 (18.92) | 81.90 (11.36)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 2 Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Physical functioning Cycle 2 Day 1 | 1.48 (9.02) | 2.22 (6.89)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Physical functioning Cycle 3 Day 28 | -2.81 (15.45) | 2.67 (5.96)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 5 Day 28: number analyzed (Participants) | 15 | 6
  EORTC QLQ-C30 Scores: Physical functioning Cycle 5 Day 28 | 1.43 (16.16) | -2.22 (5.44)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Physical functioning Cycle 8 (Week 32) | 5.45 (15.72) | -4.00 (7.60)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Physical functioning Cycle 11 Day 28 | -1.11 (6.55) | -10.00 (14.14)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Physical functioning Cycle 14 Day 28 | -1.11 (2.72) | 0.00 (9.43)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Physical functioning Cycle 17 Day 28 | 1.67 (3.33) | 0 (0)
  EORTC QLQ-C30 Scores: Physical functioning Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Physical functioning Cycle 20 Day 28 | 0 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Physical functioning Final visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Physical functioning Final visit | -4.44 (9.65) | -2.67 (7.60)
  EORTC QLQ-C30 Scores: Global health status/QoL Baseline | 61.25 (20.28) | 60.71 (7.93)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 2 Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 2 Day 1 | 2.31 (18.92) | 1.39 (8.19)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 3 Day 28: number analyzed (Participants) | 18 | 5
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 3 Day 28 | 7.89 (14.56) | 11.67 (9.50)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 5 Day 28 | 7.14 (19.84) | 0.00 (17.48)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 8 (Week 32) | 9.09 (23.41) | -8.33 (13.18)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 11 Day 28 | 1.39 (23.81) | 8.33 (11.79)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 14 Day 28 | 2.78 (21.52) | 8.33 (0)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 17 Day 28 | 10.42 (20.83) | 16.67 (0)
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Global health status/QoL Cycle 20 Day 28 | 25.00 (0) | 25.00 (0)
  EORTC QLQ-C30 Scores: Global health status/QoL Final visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Global health status/QoL Final visit | -3.33 (23.32) | 13.33 (17.28)
  EORTC QLQ-C30 Scores: Role functioning Baseline | 74.17 (28.85) | 76.19 (16.27)
  EORTC QLQ-C30 Scores: Role functioning Cycle 2 Day 1: number analyzed (Participants) | 18 | 6
  EORTC QLQ-C30 Scores: Role functioning Cycle 2 Day 1 | 7.41 (17.36) | -8.33 (17.48)
  EORTC QLQ-C30 Scores: Role functioning Cycle 3 Day 28: number analyzed (Participants) | 19 | 5
  EORTC QLQ-C30 Scores: Role functioning Cycle 3 Day 28 | 2.63 (17.80) | 0.00 (11.79)
  EORTC QLQ-C30 Scores: Role functioning Cycle 5 Day 28: number analyzed (Participants) | 14 | 6
  EORTC QLQ-C30 Scores: Role functioning Cycle 5 Day 28 | 7.14 (15.63) | -2.78 (22.15)
  EORTC QLQ-C30 Scores: Role functioning Cycle 8 (Week 32): number analyzed (Participants) | 11 | 5
  EORTC QLQ-C30 Scores: Role functioning Cycle 8 (Week 32) | 15.15 (21.67) | 0.00 (20.41)
  EORTC QLQ-C30 Scores: Role functioning Cycle 11 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Role functioning Cycle 11 Day 28 | -2.78 (19.48) | -8.33 (11.79)
  EORTC QLQ-C30 Scores: Role functioning Cycle 14 Day 28: number analyzed (Participants) | 6 | 2
  EORTC QLQ-C30 Scores: Role functioning Cycle 14 Day 28 | 5.56 (8.61) | 0 (0)
  EORTC QLQ-C30 Scores: Role functioning Cycle 17 Day 28: number analyzed (Participants) | 4 | 2
  EORTC QLQ-C30 Scores: Role functioning Cycle 17 Day 28 | 8.33 (9.62) | 0 (0)
  EORTC QLQ-C30 Scores: Role functioning Cycle 20 Day 28: number analyzed (Participants) | 1 | 1
  EORTC QLQ-C30 Scores: Role functioning Cycle 20 Day 28 | 16.67 (0) | 0 (0)
  EORTC QLQ-C30 Scores: Role functioning Final Visit: number analyzed (Participants) | 15 | 5
  EORTC QLQ-C30 Scores: Role functioning Final Visit | -13.33 (32.24) | 6.67 (9.13)

40. Secondary Outcome: Frequency Count of Participant Responses to the Patient Global Impression of Change (PGIC) Question Over Time
Description: The PGIC is a one-item measure used to assess perceived treatment benefit. Participants were asked "Since the start of the treatment you've received in this study, your polycythemia vera (PV) symptoms are: 'very much improved', 'much improved', 'minimally improved', 'no change', 'minimally worse', 'much worse', and 'very much worse'.
  The study was pre-maturely terminated by the sponsor's decision, therefore did not reach the end of study.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 28, Cycle 5 Day 28, End of Cycle 8 (Week 32), and every 3 cycles thereafter (1 cycle is 28 days) until end of study (up to 2 years)
Population: ITT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Count of Participants
Arm/Group | Ruxolitinib-Naïve Participants | Ruxolitinib-Resistant or Intolerant Participants
Number analyzed (Participants) | 20 | 7
Count of Participants
  Cycle 2, Day 1 Very Much Improved: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Very Much Improved | 0 | 0
  Cycle 2, Day 1 Much Improved: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Much Improved | 4 | 1
  Cycle 2, Day 1 Minimally Improved: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Minimally Improved | 5 | 3
  Cycle 2, Day 1 No Change: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 No Change | 6 | 1
  Cycle 2, Day 1 Minimally Worse: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Minimally Worse | 1 | 1
  Cycle 2, Day 1 Much Worse: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Much Worse | 0 | 0
  Cycle 2, Day 1 Very Much Worse: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Very Much Worse | 0 | 0
  Cycle 2, Day 1 Not Assessed: number analyzed (Participants) | 16 | 7
  Cycle 2, Day 1 Not Assessed | 0 | 1
  Cycle 3 Day 28 Very Much Improved: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Very Much Improved | 4 | 1
  Cycle 3 Day 28 Much Improved: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Much Improved | 4 | 1
  Cycle 3 Day 28 Minimally Improved: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Minimally Improved | 6 | 3
  Cycle 3 Day 28 No Change: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 No Change | 3 | 0
  Cycle 3 Day 28 Minimally Worse: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Minimally Worse | 0 | 0
  Cycle 3 Day 28 Much Worse: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Much Worse | 0 | 0
  Cycle 3 Day 28 Very Much Worse: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Very Much Worse | 0 | 0
  Cycle 3 Day 28 Not Assessed: number analyzed (Participants) | 17 | 6
  Cycle 3 Day 28 Not Assessed | 0 | 1
  Cycle 5 Day 28 Very Much Improved: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Very Much Improved | 2 | 1
  Cycle 5 Day 28 Much Improved: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Much Improved | 6 | 1
  Cycle 5 Day 28 Minimally Improved: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Minimally Improved | 2 | 4
  Cycle 5 Day 28 No Change: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 No Change | 1 | 0
  Cycle 5 Day 28 Minimally Worse: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Minimally Worse | 0 | 0
  Cycle 5 Day 28 Much Worse: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Much Worse | 0 | 0
  Cycle 5 Day 28 Very Much Worse: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Very Much Worse | 0 | 0
  Cycle 5 Day 28 Not Assessed: number analyzed (Participants) | 15 | 6
  Cycle 5 Day 28 Not Assessed | 4 | 0
  Week 32 Very Much Improved: number analyzed (Participants) | 11 | 5
  Week 32 Very Much Improved | 3 | 0
  Week 32 Much Improved: number analyzed (Participants) | 11 | 5
  Week 32 Much Improved | 3 | 1
  Week 32 Minimally Improved: number analyzed (Participants) | 11 | 5
  Week 32 Minimally Improved | 3 | 3
  Week 32 No Change: number analyzed (Participants) | 11 | 5
  Week 32 No Change | 1 | 1
  Week 32 Minimally Worse: number analyzed (Participants) | 11 | 5
  Week 32 Minimally Worse | 1 | 0
  Week 32 Much Worse: number analyzed (Participants) | 11 | 5
  Week 32 Much Worse | 0 | 0
  Week 32 Very Much Worse: number analyzed (Participants) | 11 | 5
  Week 32 Very Much Worse | 0 | 0
  Week 32 Not Assessed: number analyzed (Participants) | 11 | 5
  Week 32 Not Assessed | 0 | 0
  Cycle 11 Day 28 Very Much Improved: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Very Much Improved | 1 | 0
  Cycle 11 Day 28 Much Improved: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Much Improved | 3 | 2
  Cycle 11 Day 28 Minimally Improved: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Minimally Improved | 0 | 0
  Cycle 11 Day 28 No Change: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 No Change | 0 | 0
  Cycle 11 Day 28 Minimally Worse: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Minimally Worse | 1 | 0
  Cycle 11 Day 28 Much Worse: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Much Worse | 0 | 0
  Cycle 11 Day 28 Very Much Worse: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Very Much Worse | 0 | 0
  Cycle 11 Day 28 Not Assessed: number analyzed (Participants) | 5 | 2
  Cycle 11 Day 28 Not Assessed | 0 | 0
  Cycle 14 Day 28 Very Much Improved: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Very Much Improved | 2 | 0
  Cycle 14 Day 28 Much Improved: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Much Improved | 2 | 2
  Cycle 14 Day 28 Minimally Improved: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Minimally Improved | 0 | 0
  Cycle 14 Day 28 No change: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 No change | 1 | 0
  Cycle 14 Day 28 Minimally Worse: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Minimally Worse | 1 | 0
  Cycle 14 Day 28 Much Worse: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Much Worse | 0 | 0
  Cycle 14 Day 28 Very Much Worse: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Very Much Worse | 0 | 0
  Cycle 14 Day 28 Not Assessed: number analyzed (Participants) | 6 | 2
  Cycle 14 Day 28 Not Assessed | 0 | 0
  Cycle 17 Day 28 Very Much Improved: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Very Much Improved | 1 | 0
  Cycle 17 Day 28 Much Improved: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Much Improved | 1 | 2
  Cycle 17 Day 28 Minimally Improved: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Minimally Improved | 1 | 0
  Cycle 17 Day 28 No Change: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 No Change | 1 | 0
  Cycle 17 Day 28 Minimally Worse: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Minimally Worse | 0 | 0
  Cycle 17 Day 28 Much Worse: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Much Worse | 0 | 0
  Cycle 17 Day 28 Very Much Worse: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Very Much Worse | 0 | 0
  Cycle 17 Day 28 Not Assessed: number analyzed (Participants) | 4 | 2
  Cycle 17 Day 28 Not Assessed | 0 | 0
  Cycle 20 Day 28 Very Much Improved: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Very Much Improved | 0 | 0
  Cycle 20 Day 28 Much Improved: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Much Improved | 0 | 0
  Cycle 20 Day 28 Minimally Improved: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Minimally Improved | 1 | 0
  Cycle 20 Day 28 No Change: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 No Change | 0 | 0
  Cycle 20 Day 28 Minimally Worse: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Minimally Worse | 0 | 0
  Cycle 20 Day 28 Much Worse: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Much Worse | 0 | 0
  Cycle 20 Day 28 Very Much Worse: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Very Much Worse | 0 | 0
  Cycle 20 Day 28 Not Assessed: number analyzed (Participants) | 1 | 1
  Cycle 20 Day 28 Not Assessed | 0 | 0
  Final Visit Very Much Improved: number analyzed (Participants) | 17 | 5
  Final Visit Very Much Improved | 3 | 1
  Final Visit Much Improved: number analyzed (Participants) | 17 | 5
  Final Visit Much Improved | 3 | 3
  Final Visit Minimally Improved: number analyzed (Participants) | 17 | 5
  Final Visit Minimally Improved | 2 | 1
  Final Visit No Change: number analyzed (Participants) | 17 | 5
  Final Visit No Change | 6 | 0
  Final Visit Minimally Worse: number analyzed (Participants) | 17 | 5
  Final Visit Minimally Worse | 1 | 0
  Final Visit Much Worse: number analyzed (Participants) | 17 | 5
  Final Visit Much Worse | 0 | 0
  Final Visit Very Much Worse: number analyzed (Participants) | 17 | 5
  Final Visit Very Much Worse | 0 | 0
  Final Visit Not Assessed: number analyzed (Participants) | 17 | 5
  Final Visit Not Assessed | 2 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to end of study (up to 2 years) post initial dose or until subject discontinued. Safety follow-up: Until 28 days after the last dose of study treatment or until initiating another anti-cancer therapy.
Description: Reported: Safety Population. During the Safety Follow-up Period, non-Serious Adverse Events occurred at the 5% frequency threshold.
Groups:
- Ruxolitinib Naive-With Splenomegaly; Ruxolitinib Naive-Without Splenomegaly; Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly; Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly: Participants received 150 milligrams (mg) idasanutlin orally, once daily for 5 days, every 28 days, until treatment discontinuation or end of study (up to 2 years).
Arm/Group | Ruxolitinib Naive-With Splenomegaly | Ruxolitinib Naive-Without Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/5 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 15/15 | 5/5 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Naive-With Splenomegaly (N=15) | Ruxolitinib Naive-Without Splenomegaly (N=5) | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly (N=6) | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly (N=1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Naive-With Splenomegaly (N=15) | Ruxolitinib Naive-Without Splenomegaly (N=5) | Ruxolitinib-Resistant or Intolerant Participants With Splenomegaly (N=6) | Ruxolitinib-Resistant or Intolerant Participants Without Splenomegaly (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3) | 1 (2) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (2) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (7) | 0 (0) | 3 (5) | 1 (6)
Diarrhoea (Gastrointestinal disorders) | 11 (38) | 3 (11) | 6 (9) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (60) | 5 (15) | 6 (25) | 1 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (12) | 3 (4) | 1 (2) | 1 (1)
Asthenia (General disorders) | 2 (6) | 1 (2) | 1 (4) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (27) | 0 (0) | 4 (13) | 1 (3)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 0 (0) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 1 (5) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Solitary fibrous tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (9) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (4) | 3 (4) | 1 (1)
Migraine (Nervous system disorders) | 2 (8) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 5 (14) | 0 (0) | 0 (0) | 1 (4)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (3) | 1 (2)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03287245/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03287245/SAP_001.pdf